# STATISTICAL ANALYSIS PLAN STUDY W15-679 (STRIKE)

Version 1.0

03 April 2018

# **General Information**

| Protocol | STRIKE – Treating Patients with Early Axial Spondyloarthritis to Target – a 1<br>Year Randomized Controlled Study Taking an Intense Treatment Approach<br>Versus Routine Treatment - W15-679 |
|---|---|
| Document definition | Statistical Analysis Plan (SAP) – Version 1.0. 03 April 2018 |
| Related<br>Documents | Study Protocol, dated 30 March 2017 |
| Document owner | IST GmbH, Soldnerstrasse 1, D-68219 Mannheim |

| | | TABLE OF CONTENTS | Page |
|----|---------|-----------------------------------------------|------|
| 1. | INTROE | DUCTION | 6 |
| 2. | STUDY | OBJECTIVES | 6 |
| 3. | STUDY | DESIGN | 8 |
| | 3.1 | Overview of Study Design and Dosing Regimen | 8 |
| | 3.2 | Sample Size Calculation | |
| 4. | STATIS | TICAL CONSIDERATIONS AND ANALYTICAL PLAN | 11 |
| | 4.1 | Primary and Secondary Efficacy Parameters | 11 |
| | 4.1.1 | Primary Efficacy Parameter | |
| | 4.1.2 | Secondary Efficacy Parameters | |
| | 4.2 | Statistical and Analytical Methods | |
| | 4.2.1 | Analysis Populations | |
| | 4.2.2 | Definition of Baseline and Visit Time Windows | |
| | 4.2.3 | Patient Disposition | 21 |
| | 4.2.4 | Baseline Characteristics | |
| | 4.2.4.1 | Demographic Characteristics | 22 |
| | 4.2.4.2 | Medical and Surgical History | |
| | 4.2.4.3 | Laboratory Data | |
| | 4.2.4.4 | Prior medication | |
| | 4.2.5 | Analyses of Efficacy | 25 |
| | 4.2.5.1 | Primary Variable | |
| | 4.2.5.2 | Secondary Variables | |
| | 4.2.5.3 | Exploratory Analyses | |
| | 4.2.5.4 | Subgroup Analyses | |
| | 4.2.6 | Analyses of Safety | |
| | 4.2.6.1 | Exposure to Study Medication | |
| | 4.2.6.2 | Adverse Events | |
| | 4.2.6.3 | Laboratory Data | |
| | 4.2.6.4 | Vital Signs | |
| | 4.2.6.5 | Co-medication | |
| | 4.2.7 | Interim Analyses | 33 |
| | 4.2.8 | Protocol Violations and Deviations | |
| 5. | DATA Ç | QUALITY ASSURANCE | 34 |
| 6. | METHO | DDS OF DATA ANALYSIS AND PRESENTATION | 35 |

| | 6.1 | Analysis Data Sets | 35 |
|----|--------|--------------------|----|
| | 6.2 | SAS Output Format | 35 |
| 7. | REFERE | NCES | 36 |

# **GLOSSARY OF ABBREVIATIONS**

| AE | Adverse Event |
|---|---|
| ALT | Alanine aminostransferase |
| AS | Ankylosing Spondylitis |
| ASAS | Assessment of Spondyloarthritis International Society |
| ASAS HI | Assessment of Spondyloarthritis International Society Health Index |
| AST | Aspartate aminostransferase |
| axSpA | Axial Spondyloarthritis |
| BASDAI | Bath Ankylosing Spondylitis Disease Activity Index |
| BASFI | Bath Ankylosing Spondylitis Functional Index |
| BASMIlin | Linear Bath Ankylosing Spondylitis Metrology Index |
| CI | Confidence Interval |
| CD74 CLIP | Cluster of Differentiation 74 Class II-associated Invariant<br>Chain Peptide |
| CRF | Case Report Form |
| CRP | C-reactive Protein |
| eCRF | Electronic Case Report Form |
| EQ-5D | European Quality of Life – 5 Dimension Questionnaire |
| ESR | Erythrocyte Sedimentation Rate |
| HBc Ab | Hepatitis B core antibody |
| HBs Ab | Hepatitis B surface antibody |
| HBs Ag | Hepatitis B Surface Antigen |
| HBV | Hepatitis B virus |
| HI | Health Index |
| HIV | Human Immunodeficiency Virus |
| HLA-B27 | Human Leukocyte Antigen-B27 |
| HPF | High-power field |
| ITT | Intent to Treat |
| MASES | Maastricht Ankylosing Spondylitis Enthesitis Score |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Imaging |

# **GLOSSARY OF ABBREVIATIONS**

| NA | Not Available |
|----------------|---------------------------------------------------|
| ND | Not Done |
| NRS | Numerical Rating Scale |
| NSAID | Nonsteroidal Anti-inflammatory Drug |
| PCR | Polymerase chain reaction |
| PP | Per-protocol |
| RA | Rheumatoid Arthritis |
| RBC | Red Blood Cell |
| SI | Sacroiliac |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SI | Système International d'Unités |
| SOC | Standard of Care |
| SpA | Spondyloarthritis |
| T2T | Treat to Target |
| TAI | Total Activity Impairment |
| TB | Tuberculosis |
| TNF | Tumor Necrosis Factor |
| $TNF\alpha \\$ | Tumor Necrosis Factor Alpha |
| TWP | Total Work Productivity Impairment |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cell |
| WPAI- | Work Productivity and Activity Impairment – axSpA |
| axSpA | |

## 1. INTRODUCTION

There is an unmet medical need for the treatment of axial spondyloarthritis (axSpA). In this study, a 'treat to target' (T2T) treatment scheme escalating to combination treatment with one nonsteroidal anti-inflammatory drug (NSAID) and adalimumab (if needed) is investigated.

According to the ASAS and European League Against Rheumatism (EULAR) recommendations, NSAIDs are the first line of therapy in symptomatic patients with axSpA. Tumor necrosis factor alpha (TNF $\alpha$ )-blocking agents (TNF-blockers) are recommended in active axSpA with predominant axial manifestations if patients are still active after starting an NSAID therapy or if there are contraindication for an NSAID therapy. However, conventional DMARDs are not effective for the treatment the axial component of spondyloarthritis (SpA). In case of peripheral arthritis and/or enthesitis local glucocorticosteroid injections can be considered. Currently NSAIDs and TNF-blockers are the only effective and approved drugs for the treatment of axSpA.

Adalimumab (the TNF-blocker used in this study) was first approved for the treatment of subjects with rheumatoid arthritis (RA) in the United States (US) in December 2002 and in the European Union (EU) in September 2003. Adalimumab therapy has a well-established and well described safety profile based on extensive post-marketing experience and continued clinical trial patient exposure since the first approved indication in 2002 for rheumatoid arthritis.

Recently, similar to previous T2T recommendations for RA, T2T recommendations for the whole group of SpA including patients with axSpA and psoriatic arthritis have been developed. However, axSpA treatment targets and treatment escalation strategies have not been identified and validated in a prospective study.

Therefore, in this study an intensified T2T treatment approach comprising clearly defined treatment targets and cut-offs for treatment escalation shall be investigated in comparison to standard of care (SOC) treatment.

#### 2. STUDY OBJECTIVES

The objectives of this study are:

#### Primary objective:

The primary objective of this study is to compare a T2T intense treatment approach with a routine treatment approach (SOC) in reducing disease activity at Week 32 in patients with axSpA.

Secondary objectives are to compare a T2T intense treatment approach with SOC by assessing the following at Week 32 and Week 52:

Improvement of quality of life

- Quality of life by the European Quality of Life 5 Dimension Questionnaire (EQ-5D)
- Overall functioning by Assessment of Spondyloarthritis International Society (ASAS)
   Health Index (HI)

#### Improvement of function

• Function – Represented by the Bath Ankylosing Spondylitis (AS) Functional Index (BASFI) Numerical Rating Scale (NRS) score (0 to 10)

## Improvement of work productivity

• Work Productivity and Activity Impairment – Axial Spondyloarthritis (WPAI-axSpA)

#### Reducing inflammation

- Active inflammation as measured by magnetic resonance imaging of the sacroiliac joints and the spine (Berlin Magnetic Resonance Imaging [MRI] scores for the sacroiliac [SI] joints and spine)
- C-reactive protein (CRP)
- Erythrocyte sedimentation rate (ESR)

#### Reducing disease activity

- Disease activity as measured by Bath AS Disease Activity Index (BASDAI)
- Percentage of subjects achieving 50% improvement in BASDAI (BASDAI 50 response)
- Change from Baseline in disease activity measured by Ankylosing Spondylitis Disease Activity Score (ASDAS)
- Percentage of subjects achieving ASDAS major improvement
- Percentage of subjects achieving ASDAS clinically important improvement
- Percentage of subjects in ASDAS inactive disease (ASDAS < 1.3)
- Percentage of subjects with low disease activity (ASDAS < 2.1)
- Percentage of subjects with moderate disease activity (ASDAS  $\geq$  1.3 to  $\leq$  2.1)
- Percentage of subjects with high disease activity (ASDAS  $\geq$  2.1 to  $\leq$  3.5)
- Percentage of subjects with very high disease activity (ASDAS  $\geq$  3.5)
- Percentage of subjects achieving ASAS 20, ASAS 40, and ASAS Partial Remission
- Change from Baseline in Physician's Global Assessment of Disease Activity
- Change from Baseline in Patient's Global Assessment of Disease Activity
- Change from Baseline in Patient's Global Assessment of Pain
- Change from Baseline in Swollen Joint Count (66 joints)
- Change from Baseline in Tender Joint Count (68 joints)
- Change from Baseline in the Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
- Change from Baseline in the Dactylitis count (0-20)

- Change from Baseline in Linear Bath Ankylosing Spondylitis Metrology Index (BASMIlin)
- Anterior uveitis

Other variables to be analyzed at various time points including Week 32 and Week 52:

- ASDAS course over time
- BASDAI course over time

#### **Exploratory Objectives:**

- Serum autoantibodies against cluster of differentiation 74 class II-associated invariant chain peptide (CD74 CLIP)
- Reduction of disease progression (as measured by MRI of the sacroiliac joints and the spine)

## 3. STUDY DESIGN

## 3.1 Overview of Study Design and Dosing Regimen

This is a Phase 4, multicenter, randomized, open-label, parallel-group study comparing an intensified T2T treatment approach with SOC.

The study duration will include a 42-day Screening period, a 52-week treatment period (treatment T2T according to randomization or SOC), and – only for subjects who receive study drug Humira (adalimumab) but do not continue on commercially available Humira after the study – a 70 day follow-up phone call.

Subjects who have signed the informed consent and who fulfill all screening criteria will be randomized 1:1 to receive either treatment following an intensified T2T approach (T2T group) or treatment according to SOC (following the local practice standards) (SOC group). Study drug will only be administered to patients of the T2T group escalated to Escalation Step 2. Length of exposure will depend on individual necessity for intensifying treatment. The maximal duration of treatment with adalimumab is up to 48 weeks.

#### T2T Group (Investigational Group):

After randomization subjects are seen at Weeks 2, 4, 6, 8 and afterwards every 4 weeks up to Week 52.

Basic treatment will be started with a non-steroidal anti-inflammatory drug (NSAID). Treatment should be intensified (escalated) beginning at Week 4 if the ASDAS is  $\geq 2.1$  (escalation step 1). Treatment escalation is planned to be initiated at Week 4, if needed and further escalation is planned at Week 8, if needed (escalation step 2). However, if not required at Week 8, treatment can be escalated at every visit thereafter if the ongoing treatment is not sufficiently efficacious and the escalation step 2 has not yet been reached. Treatment escalation steps are as follows:

Basic treatment (NSAID 1): Treatment will be started with any NSAID and given for 4
weeks at full anti-inflammatory dose. If at Week 2 ASAS 20 response is not achieved,
subjects may escape early to Escalation Step 1. If the chosen NSAID cannot be continued
due to intolerance, escalation to the next escalation step is possible at any time point. If
basic treatment is well tolerated and sufficiently efficacious the subject will be continued
on this treatment.

- Escalation step 1 (NSAID 2): Treatment will be changed to a second NSAID if after 4 weeks of treatment the first NSAID is not sufficiently efficacious (ASDAS ≥ 2.1) and/or not tolerated. The second NSAID will be given for 4 weeks. Early escape is possible if after 2 weeks no ASAS 20 response is achieved. In this case treatment can be switched to escalation step 2 after 2 weeks of NSAID 2. If the chosen NSAID cannot be continued due to intolerance, escalation to the next escalation step is possible at any time point. If NSAID 2 treatment is well tolerated and sufficiently efficacious the subject will be continued on this treatment.
- Escalation step 2 (Combination with adalimumab): In case of failure of NSAID 2
   (ASDAS ≥ 2.1 after 4 weeks of NSAID 2) the treatment will be intensified by switching
   to the combination of NSAID and adalimumab 40 mg s.c. every other week (eow).
   Escalation step 2 can be initiated at Week 4 visit at the earliest if early escape is chosen
   during Basic Treatment and during NSAID 2.

#### SOC Group (Reference Group):

After randomization, subjects will receive treatment according to local practice standards. Subjects are seen at Weeks 12, 24, 32, and 52.

Figure 1. Study Design Schematic



<sup>\*</sup> Escalation schedule for the T2T intensified treatment see below.

# **Escalation in the T2T intensified treatment group**



§ Early escape after 2 wks NSAIDs intake: In case of no ASAS 20 response or intolerance switch to next escalation step (2<sup>nd</sup> NSAID/NSAID+ADA)

## 3.2 Sample Size Calculation

Based on available data from previous studies it is assumed that ASDAS inactive disease could be reached by 40% in the T2T group versus 20% in the control group. In total  $2 \times 90$  evaluable subjects are necessary to detect with 80% power an increase in ASDAS inactive disease at Week 32 from 20% in the SOC arm to 40% in the intensified T2T arm, if a two sided Fisher's exact test is applied. If the Pearson chi-square test instead of the Fisher's exact test can be applied, then only  $2 \times 83$  subjects are necessary.

Assuming that about 18% of the randomized subjects will drop out prior to Week 32 and have to be counted as non-responder the assumed ASDAS inactive disease rate will be diluted to 16.4% in the SOC arm and 32.8% in the intensified T2T arm. The necessary sample size for this scenario (intent to treat [ITT] population) is  $2 \times 109$  subjects for the chi-square test and  $2 \times 119$  subjects for the Fisher's exact test. In summary,  $2 \times 120$  subjects should be randomized.

## 4. STATISTICAL CONSIDERATIONS AND ANALYTICAL PLAN

## 4.1 Primary and Secondary Efficacy Parameters

## 4.1.1 Primary Efficacy Parameter

The primary efficacy parameter is the clinical disease activity at Week 32 measured by the ASDAS.

The ASDAS is defined as follows:

 $ASDAS_{CRP} = 0.12 \times total back pain [BASDAI question 2] + 0.110 \times global disease activity [Patient global assessment of disease activity] + 0.07 \times peripheral pain/swelling [BASDAI question 3] + 0.06 \times duration of morning stiffness [BASDAI question 6] + 0.58 \times ln(CRP [in mg/L]+1)$ 

ASDAS<sub>ESR</sub> (Alternative) =  $0.08 \times$  total back pain [BASDAI question 2] +  $0.110 \times$  global disease activity [Patient global assessment of disease activity] +  $0.09 \times$  peripheral pain/swelling [BASDAI question 3] +  $0.07 \times$  duration of morning stiffness [BASDAI question 6] +  $0.29 \times \sqrt{\text{ESR}}$  [in mm/hr]

Inactive disease is defined as ASDAS < 1.3. Low disease activity is defined as ASDAS < 2.1, moderate disease activity as ASDAS  $\geq$  1.3 to < 2.1, high disease activity as ASDAS  $\geq$  2.1 to  $\leq$  3.5, and very high disease activity as ASDAS  $\geq$  3.5. [3-7]

To follow ASAS, the evaluation of total back pain will be changed from patient's assessment of total back pain (as described in the Protocol) to result of BASDAI question 2.

No imputation will be performed for missing items, and in case of missing items no index score will be calculated.

## 4.1.2 Secondary Efficacy Parameters

Secondary efficacy parameters are:

## Quality of life by the European Quality of Life (EQ-5D)

The EQ-5D-3L is a health state utility instrument that evaluates preference for health status (utility). The 5 items in the EQ-5D-3L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 3 levels of severity (1: indicating no problem, 2: indicating some/moderate problems, 3: indicating extreme problems), and a separate VAS.

Patients' responses to the EQ-5D-3L will be combined into a unique health state using a 5-digit code with one digit from each of the 5 dimensions representing the level of severity. These EQ-5D-3L states will be converted into a single preference-weighted health utility index score by applying country-specific weights. [1]

No imputation will be performed for missing items, and in case of missing items no index score will be calculated.

#### Work Productivity and Activity Impairment – axSpA (WPAI-axSpA)

The WPAI questionnaire will be used to measure work absenteeism, work presenteeism, and daily activity impairment. The WPAI-axSpA V2.0 is the axSpA specific questionnaire that will be used in this study. The WPAI-axSpA consists of 6 questions (Q1-Q6). Respondents are asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity:

- % Presenteeism percentage of impairment while working due to health problem: 100\*Q5/10
- % Absenteeism percentage of work time missed due to health problem: 100\*Q2/(Q2+Q4)
- % Total work productivity impairment (TWP) percentage of overall work impairment due to health problem: 100\*{Q2/(Q2+Q4) + [Q4/(Q2+Q4)]\* Q5/10}
- % Total activity impairment (TAI) percentage of general (non-work) activity impairment due to health problem: 100\*Q6/10

The four scores will be derived according to the WPAI-SHP scoring manual [2] using the following coding rules for contradictory or missing information:

- If employed = YES or employed = NO or missing and hours missed or worked > 0, then employed. If employed = missing and hours missed and worked = 0, then not employed.
- If hours worked = 0, then productivity while at work is not applicable.
- A score will be set to missing if one or more of the items Q1-6 that are needed for the calculation of the score are missing. No imputation will be performed for missing items.

• Someone who missed all work hours due to health is 100% impaired.

#### **Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)**

The subject will assess his/her disease activity in answering 6 questions pertaining to symptoms experienced by the subject during the past week on a numerical rating scales (NRS, 0 = None to 10 = 0 to 5 = 1h to 10 = 2 or more h). The score is defined as follows:

```
BASDAI Score = 0.2 \times (\text{Item } 1 + \text{Item } 2 + \text{Item } 3 + \text{Item } 4 + 0.5 \times \text{Item } 5 + 0.5 \times \text{Item } 6)
```

A major clinical response will be defined as a 50% improvement or more of the initial BASDAI (BASDAI 50). [8, 9]No imputation will be performed for missing items, and in case of missing items no score will be calculated.

## **Bath Ankylosing Spondylitis Functional Index (BASFI)**

The subject will assess his/her ability of ten selected activities for the past week using a NRS (0= easy to 10=Impossible). The BASFI is the mean of these 10 item scores.[8]

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

## Linear Bath Ankylosing Spondylitis Metrology Index (BASMI<sub>lin</sub>)

The BASMI will be conducted at the designated study visits to evaluate spinal mobility in a subject. The five assessments are scored as follows:

| • | Lateral lumbar flexion (mean right/left) | (21.1 cm - RESULT)/2.1 cm |
|---|-------------------------------------------|---------------------------|
| • | Tragus to wall distance (mean right/left) | (RESULT - 8 cm)/3 cm |
| • | Lumbar flexion (modified Schober) | (7.4 cm - RESULT)/0.7 cm |
| • | Maximal intermalleolar distance | (124.5 cm - RESULT)/10 cm |
| • | Cervical rotation angle (mean right/left) | (89.3° - RESULT)/8.5° |

The mean score of the five assessments gives the BASMI linear result (0-10). [8]

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### Magnetic Resonance Imaging (MRI) of the Spine and Sacroiliac Joints

All subjects will have a MRI evaluation of the sacroiliac (SI) joints as well as the cervical, thoracic and lumbar regions of the spine at screening and the last visit (at week 52 visit or – in case of early discontinuation – the discontinuation visit). Images will be sent to the central imaging vendor designated by the Sponsor. Images will be scored for inflammatory lesions and chronic structural changes in the spine and the sacroiliac joints using a modified version of the Berlin MRI score. [11] For this purpose, each SI joint will be divided into four quadrants and the

spine into 23 vertebral units which will be rated according to Table 1. Summing up the gradings yields the following scores:

- Sacroiliac joints
  - o Active inflammation (0-24)
  - o Erosion (0-24)
  - o Fatty deposition (0-24)
  - o Sclerosis (0-2)
  - o Ankylosis (0-2)
- Spine
  - o Active Inflammation (0-69)
  - o Erosion (0-23)
  - o Fatty deposition (0-69)
  - o Bone proliferation (0-69)
  - o Activity in facet joints (0-23)
  - o Activity in Proc. spinosus (0-23)
  - o Activity of soft tissue in posterior spinal sites (0-23)

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

Table 1 Berlin Magnetic Resonance Imaging (MRI) Score for the Spine and the Sacroiliac Joints

| | Grade 0 | Grade 1 | Grade 2 | Grade 3 |
|---|---|---|---|---|
| Sacroiliac joints | | | | |
| Active inflammation (BMO of quadrant area) | Absent | Up to 33% of the quadrant area | 33% – 66% | %99 < |
| Erosions (per quadrant) | Absent | Minor (one to two erosions) | Moderate (three to five single erosions | Multiple (confluent erosions) |
| Fatty bone marrow deposition (per quadrant) | Absent | < 33% | 3366% | %99< |
| Sclerosis (per joint) | Absent | Present | ŀ | ! |
| Ankylosis (per joint) | Absent | Present | 1 | ŀ |
| Spine | | | | |
| Active Inflammation (BMO of VU area) | Absent | < 33% of VU area | 33% – 66% | %99 < |
| Erosions (% of the bone surface per VU) | Absent | present | | |
| Fatty bone marrow deposition (per VU) | Absent | <33% | 33% – 66% | %99 < |
| Bone proliferation (per VU) | Absent | Syndesmophytes without bridging | Bridging syndesmophytes | Transdiscal ankylosis |
| Activity in facet joints (right and/or left) | Absent | present | | I |
| Activity in Proc. spinosus | Absent | present | | |
| Activity of soft tissue in posterior spinal sites | Absent | present | | |

BMO = bone marrow edema; VU = vertebral unit

#### **Assessment of Disease Activity and Pain**

NRSs will be used to assess:

- Physician's global assessment of disease activity
- Patient's global assessment of disease activity
- Patient's global assessment of pain
- Patient's assessment of nocturnal back pain within the last week
- Patient's assessment of total back pain within the last week.

The left end of the NRS (0) signifies the absence of symptoms and the right end (10) signifies maximum activity or pain.

## Assessment of Spondyloarthritis International Society (ASAS) Health Index (HI)

The ASAS HI will assess the overall functioning of each subject. The responses to the 17 dichotomous items can be summed up to give a total score ranging from 0 to 17 - with a lower score indicating a better and a higher score indicating an inferior health status.[10]

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### ASAS 20, ASAS 40, and ASAS Partial Remission

The ASAS response criteria are defined as follows [6]:

- ASAS20 response: improvement of  $\geq 20\%$  and absolute improvement of  $\geq 1$  unit (on a scale of 0 to 10) from Baseline in  $\geq 3$  of the following 4 domains, with no deterioration in the remaining domain (defined as a worsening of  $\geq 20\%$  and a net worsening of  $\geq 1$  unit)
  - Patient's Global Assessment Represented by the PTGA-disease activity NRS score (0 to 10)
  - o Pain Represented by the patient's assessment of total back pain NRS score (0 to 10)
  - o Function Represented by the BASFI NRS score (0 to 10)
  - o Inflammation Represented by the mean of the 2 morning stiffness-related BASDAI NRS scores (mean of items 5 and 6 of the BASDAI [0 to 10])
- ASAS40 response: improvement of  $\geq 40\%$  and absolute improvement of  $\geq 2$  units (on a scale of 0 to 10) from Baseline in  $\geq 3$  of the 4 domains above in ASAS20 with no deterioration at all in the potential remaining domain
- ASAS partial remission: absolute score of ≤ 2 units for each of the 4 domains identified above in ASAS20

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)

At the designated study visits the presence or absence of enthesitis at 13 different sites will be assessed. All sites are scored as 0 (absent) or 1 (present). The MASES is the sum of all site scores (from 0 to 13). [8]

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### Swollen and tender joint counts

An assessment of 68 joints will be done by physical examination at the designated study visits. The joints will be examined for tenderness (score: 0-68) and swelling (score: 0-66). The joints to be examined for swelling are the same as those examined for tenderness, except the hip joints are excluded. Enthesitis is not part of the swollen joint assessment.

No imputation will be performed for missing items, and in case of missing items or joint replacements no score will be calculated.

#### **Dactylitis counts**

Evaluation for dactlyitis will be conducted at the designated study visits to assess the presence or absence of dactylitis in all 20 of the subjects' digits (score: 0-20).

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### **Anterior uveitis**

At the screening visit a detailed medical history of anterior uveitis, as confirmed by an ophthalmologist, will be documented. At baseline and all subsequent visits, new onsets of uveitis (right, left or both) and/or the number of flares since last visit will be documented.

No imputation will be performed for missing items, and in case of missing items no score will be calculated.

#### **Laboratory parameters - exploratory and efficacy analyses**

The following laboratory parameters will be assessed: C-reactive protein (CRP [mg/L]) and erythrocyte sedimentation rate (ESR [mm/h (1st hour)]). Exploratory analysis of CD74CLIP will not be performed.

For further details on the assessment of serum autoantibodies against CD74 CLIP, CRP and ESR please refer to Section 4.2.5.3.

# 4.2 Statistical and Analytical Methods

## 4.2.1 Analysis Populations

Subjects are screened to ensure they meet all inclusion criteria and none of the exclusion criteria mentioned below at both Screening and Baseline Visits.

#### Main Inclusion:

- 1. Subjects must have signed written informed consent before starting any study-related assessments or procedures.
- 2. Diagnosis of axSpA (either ankylosing spondylitis or non-radiographic axSpA) and fulfilling the ASAS classification criteria for axSpA.
- 3. Subjects aged  $\geq$  18 years.
- 4. Disease duration < 5 years.
- Subjects must have a baseline disease activity as defined by having an ASDAS ≥ 2.1 or a BASDAI ≥ 4.
- 6. Subjects must be either NSAID-naïve or had not been treated with the maximal recommended dose during the last 2 weeks prior to the Baseline Visit.
- 7. Subjects must be disease-modifying anti-rheumatic drug (DMARD)-naïve except for methotrexate (MTX), sulfasalazine (SSZ), azathioprine (AZA), and 6-mercaptopurine (6-MP).
- 8. Subjects must never have failed a NSAID taken at maximal recommended dose for 2 weeks or more.
- 9. If female, subject must be either postmenopausal, OR permanently surgically sterile OR for Women of Childbearing Potential practicing at least one protocol specified method of birth control, starting at Study Day 1 through at least 150 days after the last dose of study drug.
  - If the male subject is sexually active with female partner(s) of childbearing potential, he must agree, from Study Day 1 through 20 weeks after the last dose of study drug, to practice the protocol specified contraception.
- 10. Females of childbearing potential must have a negative serum pregnancy test result at Screening, and a negative urine pregnancy test at Baseline Visit.
  - Females of non-childbearing potential (either postmenopausal or permanently surgically sterile as defined above) at Screening do not require pregnancy testing.
- 11. Subject is judged to be in good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, and a 12-lead ECG performed at Screening.
- 12. Subjects must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections.

13. Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.

#### Main Exclusion:

- 1. Contraindications for NSAIDs or Tumor Necrosis Factor (TNF) blocker according to local labeling.
- 2. Subject has a medical condition precluding an MRI (e.g., magnetic activated implanted devices cardiac pace-maker, insulin pump, neurostimulators, etc. and metallic devices or fragments in the body).
- 3. Subject has active inflammatory bowel disease.
- 4. Prior exposure to any anti-TNF therapy; any biologic therapy with a potential therapeutic impact on SpA, or subject has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half-lives (whichever is longer) of the drug prior to the Baseline Visit.
- 5. If entering the study on concomitant NSAIDs, subjects taking the maximal recommended dose during the last 2 weeks prior to the Baseline Visit or have failed or developed intolerance to a NSAID taken at maximal recommended dose for 2 weeks or more at any time.
- 6. Subject on opioid analgesics or use of marijuana within 14 days prior to the Baseline Visit.
- 7. If entering the study on concomitant oral corticosteroids, subject has not been on stable dose of prednisone (≤ 10 mg per day), or oral corticosteroid equivalents, for at least 14 days prior to the Baseline Visit.
- 8. Subject has been treated with intra-articular joint injection(s) or spinal/paraspinal injection(s) of corticosteroids in the preceding 28 days prior to the Baseline Visit.
- 9. Subject has undergone spinal surgery within 2 months prior to Baseline or subject has been diagnosed with a spinal condition that may interfere with study assessments (i.e., disc herniation, degenerative spine disease, etc.) in the opinion of the investigator.
- 10. Subject has a history of fibromyalgia or inflammatory arthritis of a different etiology other than SpA (e.g., rheumatoid arthritis, systemic lupus erythematosus, polyarticular or systemic juvenile idiopathic arthritis).
- 11. Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline Visit or oral anti-infectives within 14 days prior to the Baseline Visit.
- 12. Known hypersensitivity to adalimum b or its excipients as stated in the label.
- 13. Known intolerance of NSAID treatment that does not allow use of at least two different NSAIDs at full anti-inflammatory dose.
- 14. History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.

- 15. History of invasive infection (e.g., listeriosis and histoplasmosis), human immunodeficiency virus (HIV).
- 16. Subjects with any active viral infection that based on the investigator's clinical assessment, makes the subject an unsuitable candidate for the study.
- 17. Hepatitis B: Hepatitis B surface antigen (HBs Ag) positive (+) or detected sensitivity on the hepatitis B virus (HBV)-DNA polymerase chain reaction (PCR) qualitative test for hepatitis B core antibody (HBc Ab)/hepatitis B surface antibody (HBs Ab) positive subjects.
- 18. Chronic recurring infections or active TB.
- 19. History of moderate to severe congestive heart failure (New York Heart Association [NYHA] class III or IV), recent cerebrovascular accident and any other condition which would put the subject at risk by participation in the study.
- 20. Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.
- 21. Positive pregnancy test at Screening or Baseline.
- 22. Female subject who is pregnant, breastfeeding or is considering becoming pregnant during the study or for approximately 150 days after the last dose of study drug.
- 23. Male subject who is considering fathering a child or donating sperm during the study or for approximately 150 days after the last dose of study drug.
- 24. Clinically significant abnormal screening laboratory results as evaluated by the Investigator.
- 25. History of clinically significant drug or alcohol abuse in the last 12 months.
- 26. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
- 27. Any vulnerable subject (e.g., person kept in detention, or dependent from the Sponsor, Investigator or study site)

**Enrolled population** is defined as all patients who signed written informed consent.

**Intent-to-treat analysis (ITT) population** is defined as all patients enrolled who were randomized.

**Safety analysis (SP) population** is defined all patients enrolled who were randomized and received treatment for axSpA after randomization.

**Per-protocol (PP) population** is defined as all patients of the ITT population who have sufficient data regarding the primary efficacy endpoint (clinical disease activity at Week 32) and did not meet any major protocol violation.

## 4.2.2 Definition of Baseline and Visit Time Windows

For each subject, study day 1 is defined as the day of randomization. For baseline analyses the last available value prior to or on the day of randomization will be used.

Subjects are allowed a visit window of  $\pm$  7 days for all study visits (after baseline).

If a subject has an out of window visit, the next visit should occur as originally scheduled based on the date of the baseline visit.

In subjects of the T2T group, HBV screening, TB screening and chest X-ray (CXR) will be performed before Escalation Step 2 is initiated (before adalimumab is administered).

If a subject is diagnosed with latent TB the subject has to undergo a minimum of 1 month of anti-TB prophylaxis before Escalation Step 2 can be initiated. In this case the time until the next visit will be counted from the start of adalimumab; e.g., if a subject starts TB prophylaxis at Week 8 visit and initiates Escalation Step 2 after receiving 2 months of prophylaxis, i.e., 16 weeks after Baseline, the next visit (nominal Week 12 visit) will be postponed by these 2 months (to 20 weeks after Baseline). All subsequent visits will be postponed accordingly, e.g., Week 16 visit to 24 weeks after Baseline.

If a subject is diagnosed with active hepatitis B the subject is not eligible to receive adalimumab and should discontinue from the study.

## 4.2.3 Patient Disposition

The absolute and relative numbers of the patients enrolled [rescreened patients are only counted once], the patients in the ITT and the patients in the SP will be displayed. The number of patients in the PP will not be displayed because the study was stopped prematurely by the sponsor. However, the number of patients of the SP who are treated for axSpA after randomization but meet at least one major protocol violation will be displayed, including the major protocol violations. Major protocol violations will be identified by an expert with the help of data listings. (See also section 4.2.8) Multiple violations could be reported per patient.

Furthermore the absolute and relative numbers of the patients completing the treatment phase and the reason why not by frequency (i.e. termination of study by sponsor, adverse event(s), failure to return, pregnancy, insufficient therapeutic response, withdrawn consent, death, other [including specifications will be displayed last]) will be displayed. Multiple reasons could be reported per patient.

Information about patient disposition will be listed as well.

An overview of tables and listings is given in Table 2.

#### 4.2.4 Baseline Characteristics

Demographic and baseline characteristics will be summarized for SP in total and by treatment groups. The number of observations, mean, standard deviation, median, quartiles, minimum and maximum will be summarized for continuous variables. Discrete variables will be summarized via counts and percentages.

All baseline characteristics will be listed. An overview of listings and tables is given in Table 2.

## 4.2.4.1 Demographic Characteristics

The following demographic characteristics will be summarized:

- Sex (Male, Female)
- Age at randomization [years], flooring the difference between date of randomization and date of birth divided by 365.25 [The year of birth is reported only, so the date of will be completed via 30th June.]
- Height [cm]
- Weight [kg]
- BMI [kg/sqm]

The last value up to and including study day 1 will be displayed.

## 4.2.4.2 Medical and Surgical History

The following variables will be summarized:

- History of Tuberculosis (TB)
  - o Past TB infection (Yes, No, Unknown)
  - High TB risk (Yes, No)
  - Former BCG vaccination (Yes, No, Unknown)
- Medical History for axSpA
  - o Uveitis (Never, Former, Current, Unknown)
  - o Inflammatory bowel disease (Never, Former, Current, Unknown)
  - o Psoriasis (Never, Former, Current, Unknown)
  - Other features of spondyloarthritis (Inflammatory back pain, Arthritis (past), Heel enthesitis (past), Good prior response to NSAIDs, Family history of SpA)
- Surgical History for axSpA
  - o History of spinal surgery for axSpA (Yes, No)
  - o History of joint replacement for axSpA (Yes, No)
  - History of surgery for axSpA (Yes, No)
  - History of arthroscopy for axSpA (Yes, No)
  - o Other medical history (Yes, No)

The last value up to and including study day 1 will be displayed.

## 4.2.4.3 Laboratory Data

The following clinical chemistry and hematology laboratory parameters will be summarized:

- Creatinine [micromol/L]
- Total bilirubin [micromol/L]
- Albumin [g/L]
- Aspartate aminostransferase [AST in U/L]
- Alanine aminostransferase [ALT in U/L]
- Glucose [mmol/L]
- Hematocrit [ratio]
- Hemoglobin [g/L]
- Red Blood Cell Count [RBC in 10\*\*12/L]
- White Blood Cell Count [WBC in 10\*\*9/L]
- Neutrophils [10\*\*9/L]
- Bands [10\*\*9/L]
- Lymphocytes [10\*\*9/L]
- Monocytes [10\*\*9/L]
- Basophils [10\*\*9/L]
- Eosinophils [10\*\*9/L]
- Platelets [10\*\*9/L]

The following parameters of macroscopic urinalysis will be summarized:

- Specific Gravity (1.005, 1.010, 1.015, 1.020, 1.025, 1.030, NA/ND)
- Ketones (Negative, Trace, +, ++, +++, NA/ND)
- Protein (Negative, Trace, +, ++, +++, ++++, NA/ND)
- Glucose (Negative, Trace, +, ++, +++, NA/ND)
- pH (4.5, 5, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, NA/ND)
- Nitrite (Negative, Positive, NA/ND)
- Blood (Negative, Trace, +, ++, +++, ++++, NA/ND)

The following parameters of microscopic urinalysis will be summarized:

- Leucocytes [number / HPF]
- Erythrocytes [number / HPF]
- Dysmorphic erythrocytes [number / HPF]
- Epithelial cells [number / HPF]
- Bacteria [number / HPF]
- Yeasts [number / HPF]
- Casts [number / HPF]
- Crystal [number / HPF]

Microscopic Urinalysis is performed if the dipstic results of macroscopic urinalysis show protein, ketones or blood greater than negative or glucose greater than normal.

The following other parameters will be summarized:

- ESR [mm/h (1st hour)]
- CRP [mg/L]
- Anti-dsDNA Antibodies (Negative, Positive)
- HLA-B27 (Negative, Positive)
- HBsAg (Negative, Positive)
- HBsAb (Negative, Positive) in patients with HBsAg negative
- HBcAb (Negative, Positive) in patients with HBsAg negative
- HBV DNA PCR (Below detection sensitivity, Meeting/exceeding detection sensitivity) in patients with HBsAg negative, HBsAb negative, and HBcAb Total positive

The last value up to and including study day 1 will be displayed. For conversion factors see 4.2.6.3.

## 4.2.4.4 Prior medication

Treatments, surgical and medical procedures will be coded by AbbVie assigning appropriate preferred terms. The absolute and relative numbers of patients taking prior drug for axSpA and other prior drugs will be displayed. The drugs will be displayed via preferred term.

The medication started prior to study day 1 will be displayed.

## 4.2.5 Analyses of Efficacy

All variables will be listed. An overview of listings, figures and tables is given in Table 2.

## 4.2.5.1 Primary Variable

ASDAS will be plotted over time by subject and treatment group for the SP. The limits 1.3, 2.1 and 3.5 will be displayed as well. No non-responder imputation or LOCF will be applied and no statistical tests and no sensitivity analysis will be performed because the study was terminated prematurely by the sponsor.

## 4.2.5.2 Secondary Variables

All secondary variables, except for CD74 CLIP (see below) will be listed only, since the study was terminated prematurely by the sponsor.

## 4.2.5.3 Exploratory Analyses

No exploratory analyses will be performed because the study was terminated prematurely by the sponsor. CD74 CLIP will not be presented as readouts have not been performed. However, data on CRP and ESR, as well as data of the MRIs, will be presented as part of the Safety Analysis, see Section 4.2.6.

## 4.2.5.4 Subgroup Analyses

No subgroup analyses will be performed.

## 4.2.6 Analyses of Safety

All variables will be listed. An overview of listings, figures and tables is given in Table 2.

# 4.2.6.1 Exposure to Study Medication

All medications taken will be listed only because the study was terminated prematurely by the sponsor.

#### 4.2.6.2 Adverse Events

Adverse events (AEs) are coded by IST GmbH. A treatment-emergent adverse event is defined as AE that starts either on or after randomization or is related to study treatment. AEs will be displayed for the SP in total and by treatment group.

An overview of the number of patients with at least one of the following AEs is given:

- AE
- Malignancy, i.e. AEs fulfilling criteria for malignancy and the patient is <=30 years at time of onset of AE
- Serious AEs (SAEs)
- Life-threatening AEs
- AEs leading to death

- AEs leading to hospitalization
- Important medical event requiring medical or surgical intervention to prevent serious outcome
- AEs leading to persistent or significant disability/incapacity
- AEs leading to congenital anomalies
- AEs possibly related to HUMIRA
- AEs leading to withdrawal of HUMIRA
- AEs leading to interruption of HUMIRA
- AEs leading to start of co-medication or therapy
- AEs leading to discontinuation of co-medication or therapy
- AEs leading to study discontinuation

Furthermore, treatment-emergent AEs will be summarized via system organ class (SOC) and preferred term once overall and once by severity.

In addition, non-serious AEs will be summarized. Here, only preferred terms are taken into account that occurred at a frequency of >=5% in any treatment group.

Serious AEs, AEs leading to death, AEs leading to hospitalization, AEs possibly related to HUMIRA, AEs leading to permanent withdrawal from HUMIRA, and AEs leading to interruption of HUMIRA intake will be listed only.

## 4.2.6.3 Laboratory Data

The following clinical hematology laboratory parameters will be plotted over time by subject and treatment group for the SP:

- Hematocrit [ratio]
- Hemoglobin [g/L]
- Red Blood Cell Count [RBC in [10\*\*12/L]]
- White Blood Cell Count [WBC in [10\*\*9/L]]
- Neutrophils [10\*\*9/L]
- Bands [10\*\*9/L]
- Lymphocytes [10\*\*9/L]
- Monocytes [10\*\*9/L]
- Basophils [10\*\*9/L]
- Eosinophils [10\*\*9/L]
- Platelets [10\*\*9/L]

The following clinical chemistry laboratory parameters will be plotted over time by subject and treatment group for the SP:

- Creatinine [micromol/L]
- Total Bilirubin [micromol/L]
- Total Bilirubin / ULN
- Albumin [g/L]
- AST [U/L]
- AST / ULN
- ALT [U/L]
- ALT / ULN
- Glucose [mmol/L]

Furthermore, ESR [mm/h (1st hour)] and CRP [mg/L] will be plotted over time by subject and treatment group for the SP.

The following parameters of microscopic urinalysis will be plotted over time by subject and treatment group for the SP:

- Leucocytes [number / HPF]
- Erythrocytes [number / HPF]
- Dysmorphic erythrocytes [number / HPF]
- Epithelial cells [number / HPF]
- Bacteria [number / HPF]
- Yeasts [number / HPF]
- Casts [number / HPF]
- Crystal [number / HPF]

Microscopic Urinalysis is performed if the dipstic results of macroscopic urinalysis show protein, ketones or blood greater than negative or glucose greater than normal.

Absolute and relative number of patients over time will be displayed for parameters of macroscopic urinalysis and other laboratory parameters. The last value up to and including the relevant visit (as defined in section 4.2.2) will be displayed.

The following parameters of macroscopic urinalysis will be summarized:

- Specific Gravity (1.005, 1.010, 1.015, 1.020, 1.025, 1.030, NA/ND)
- Ketones (Negative, Trace, +, ++, +++, ++++, NA/ND)
- Protein (Negative, Trace, +, ++, +++, ++++, NA/ND)

- Glucose (Negative, Trace, +, ++, +++, ++++, NA/ND)
- pH (4.5, 5, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, NA/ND)
- Nitrite (Negative, Positive, NA/ND)
- Blood (Negative, Trace, +, ++, +++, ++++, NA/ND)

The following conversion factors will be used:

| Parameter | In | То | <b>Conversion factor</b> |
|-----------------|------------|------------|--------------------------|
| Hematocrit | % | ratio | 0.01 |
| Hemoglobin | mmol/L | g/L | 64.5 |
| Creatinine | mg/L | micromol/L | 8.84 |
| | mg/dL | | 88.4 |
| Total Bilirubin | mg/dL | micromol/L | 17.1 |
| Albumin | g/dL | g/L | 10 |
| AST | microkat/L | U/L | 59.88 |
| ALT | microkat/L | U/L | 59.88 |
| Glucose | mg/dL | mmol/L | 0.0555 |
| | g/L | | 5.55 |
| CRP | mg/dL | mg/L | 10 |

# 4.2.6.4 Vital Signs

The following parameters will be plotted over time by subject and treatment group for the SP:

- Systolic blood pressure [mmHg]
- Diastolic blood pressure [mmHg]
- Pulse [bpm]
- Respiratory rate [breath per minute]
- Body temperature [°C]
- BMI [kg/sqm]

## 4.2.6.5 Co-medication

Treatments, surgical and medical procedures will be coded by AbbVie assigning appropriate preferred terms. Concomitant medications are defined as all medication except medication for axSpA received after day one. The absolute and relative numbers of patients taking comedications will be displayed for SP overall and by treatment group. The drugs will be displayed via preferred term.

**Table 2** Overview of Outputs

| Output Title | Output Short<br>Name | Analysis Population |
|---|---|---|
| Tables and figures | | |
| Patient Disposition by Treatment Group - EP | tdis_t_ep | Enrolled population |
| Reasons for Premature Termination of the Treatment Phase by Treatment group - SP | tps_t_SP | Safety population |
| Demographic Characteristics by Treatment<br>Group – SP | tdm_t_sp | Safety population |
| Medical and Surgical History at Baseline by<br>Treatment Group – SP | tmsh_t_sp | Safety population |
| Chemistry and Hematology Laboratory<br>Variables at Baseline by Treatment Group – SP | tchl_t_sp | Safety population |
| Macroscopic Urinalysis Laboratory Variables at Baseline by Treatment Group – SP | tmaul_t_sp | Safety population |
| Microscopic Urinalysis Laboratory Variables at Baseline by Treatment Group – SP | tmiul_t_sp | Safety population |
| Other Laboratory Variables at Baseline by Treatment Group – SP | totl_t_sp | Safety population |
| Prior Medication by Treatment Group - SP | tpm_t_sp | Safety population |
| Ankylosing Spondylitis Disease Activity Score (ASDAS <sub>CRP</sub> ) by Treatment Group - SP | fasdascrp_t_sp | Safety population |
| Ankylosing Spondylitis Disease Activity Score (ASDAS <sub>ESR</sub> ) by Treatment Group - SP | fasdasesr_t_sp | Safety population |
| Overview of Treatment-emergent Adverse<br>Events by Treatment Group - SP | toae_t_sp | Safety population |
| Treatment-emergent Adverse Events by Treatment Group - SP | tae_t_sp | Safety population |
| Treatment-emergent Adverse Events by Severity and Treatment Group - SP | taes_t_sp | Safety population |
| Treatment-emergent Non-serious Adverse<br>Events by Treatment Group - SP | tnsae_t_sp | Safety population |
| Laboratory Hematology by Treatment Group – SP | flh_tc_sp | Safety population |

| Output Title | Output Short<br>Name | Analysis Population |
|---|---|---|
| Laboratory Clinical Chemistry by Treatment<br>Group – SP | flc_t_sp | Safety population |
| Laboratory Microscopic Urinalysis by Treatment<br>Group – SP | flmu_t_sp | Safety population |
| Vital Signs by Treatment Group - SP | fvs_t_sp | Safety population |
| Laboratory Macroscopic Urinalysis by<br>Treatment Group – SP | tlmu_t_s | Safety population |
| Other Laboratory Tests by Treatment Group - SP | flo_t_s | Safety population |
| Concomitant Medication by Treatment Group - SP | tcmd_t_sp | Safety population |
| Glossary of System Organ Class, MedDRA<br>Preferred Terms and Verbatim Terms for<br>Adverse Events or Diseases | tgae | - |
| Glossary of Preferred Terms and Verbatim<br>Terms for Concomitant Medication | tgcom | - |
| Listings | | |
| Patient Disposition | ldis_en | Enrolled population |
| Inclusion and Exclusion Criteria | lie_en | Enrolled population |
| Baseline Demographic Characteristics | ldm_en | Enrolled population |
| Medical and Surgical History: Tobacco or Alcohol Use | ltau_en | Enrolled population |
| Medical and Surgical History: Axial Spondyloarthritis and Other History | lhao_en | Enrolled population |
| Prior Medication for axSpA | lpma_en | Enrolled population |
| All Other Prior Medication | lopm_en | Enrolled population |
| Treatment Exposure | lte_en | Enrolled population |

| Output Title | Output Short<br>Name | Analysis Population |
|---|---|---|
| Concomitant Medication | lcom_en | Enrolled population |
| Adverse Events | lae_en | Enrolled population |
| Malignancy | lmae_en | Enrolled population |
| Serious Adverse Events | lsae_en | Enrolled population |
| Adverse Events Leading to Death | laed_en | Enrolled population |
| Adverse Events Leading to Hospitalization | laeh_en | Enrolled population |
| Adverse Events Possibly Related to HUMIRA | laer_en | Enrolled population |
| Adverse Events Leading to Permanent Withdrawal from HUMIRA | laew_en | Enrolled population |
| Adverse Events Leading to Interruption of HUMIRA Intake | laei_en | Enrolled population |
| Pregnancy Test | lpt_en | Enrolled population |
| Laboratory Clinical Chemistry | llc_en | Enrolled population |
| Laboratory Hematology | llh_en | Enrolled population |
| Microscopic Urinalysis | lmiu_en | Enrolled population |
| Macroscopic Urinalysis | lmau_en | Enrolled population |
| ESR/CRP | lec_en | Enrolled population |
| Hepatitis B Testing | lhb_en | Enrolled population |
| Vital Signs/ Weight | lvs_en | Enrolled population |
| Dactylitis | lda_en | Enrolled population |
| Anterior Uveitis | lau_en | Enrolled population |
| Physical Examinations | lpe_en | Enrolled population |

| Output Title | Output Short<br>Name | Analysis Population |
|---|---|---|
| ECG | lecg_en | Enrolled population |
| Tuberculosis | ltb_en | Enrolled population |
| Chest X-Ray | lxr_en | Enrolled population |
| Ankylosing Spondylitis Disease Activity Score (ASDAS) | lasd_en | Enrolled population |
| Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | lbas_en | Enrolled population |
| Maastricht Ankylosing Spondylitis Enthesitis<br>Score (MASES) | lmas_en | Enrolled population |
| ASAS Health Index (HI) | lahi_en | Enrolled population |
| ASAS20, ASAS40 and ASAS Partial remission | lrc_en | Enrolled population |
| Bath Ankylosing Spondylitis Functional Index (BASFI) | lbasfi_en | Enrolled population |
| Bath Ankylosing Spondylitis Metrology Index (BASMI lin) | lbasmi_en | Enrolled population |
| EQ-5D | lq_en | Enrolled population |
| WPAI-axSpA | lwp_en | Enrolled population |
| Physician's/Patient's Assessment, NRS | lpa_en | Enrolled population |
| Baseline MRI with Investigator Assessments | lmribl_en | Enrolled population |
| Berlin MRI Score for MRI of Sacroiliac Joint | lbj_en | Enrolled population |
| Berlin MRI Score for MRI of Spine | lbs_en | Enrolled population |
| Tender and Swollen Joints | lts_en | Enrolled population |

The layouts of the tables mentioned above are provided in Part II of the SAP (Table Shells).

# 4.2.7 Interim Analyses

No interim analysis is planned for this study.

#### 4.2.8 Protocol Violations and Deviations

AbbVie does not allow intentional/prospective deviations from the protocol. The Principal Investigator is responsible for complying with all protocol requirements, and applicable global and local laws regarding protocol deviations. If a protocol deviation occurs (or is identified) after a subject has been enrolled, the Principal Investigator is responsible for notifying IEC/IRB regulatory authorities (as applicable), and their assigned CRO Clinical Monitor or the responsible AbbVie Clinical Monitors.

Such contact must be made as soon as possible to permit a review by AbbVie to determine the impact of the deviation on the subject and/or the study.

For the purposes of this protocol, reportable deviations are defined as:

- Subject entered into the study even though she/he did not satisfy entry criteria
- Subject who developed withdrawal criteria during the study and was not withdrawn
- Subject who received wrong treatment or incorrect dose
- Subject who received excluded or prohibited concomitant treatment

A subject may withdraw from the study at any time. The investigator may discontinue any subject's participation prematurely for any reason, including an adverse event, safety concerns or failure to comply with the protocol.

## 5. DATA QUALITY ASSURANCE

Computer logic and manual checks will be created to identify items such as inconsistent study dates. Any necessary corrections will be made to the eCRF.

An Investigator's Meeting will be held with AbbVie personnel, the investigators and their study coordinators and the Monitors for the study. This meeting will include a detailed discussion of the scientific rational, protocol, performance of study procedures, eCRF and Subject Diary and log completion, Imaging requirement, and specimen collection methods. In addition to or instead of the Investigator's Meeting, the study personnel at each site may be trained on the study procedures by a Monitor at a study initiation visit and will be given an eCRF completion guideline for reference.

The CRO Monitors will monitor each site throughout the study. Source document review will be performed against entries in the eCRF database and a quality assurance check will be performed to ensure that the investigator is complying with the protocol and regulations.

All central laboratory results will be electronically transferred from the central laboratory to the study database.

A review of the data will be conducted by a physician and clinical review team at AbbVie as specified in the safety review plan.

All statistical programs employed in the analysis and reporting of the data will be validated according the standard operating procedures of IST and results will be checked for plausibility.

## 6. METHODS OF DATA ANALYSIS AND PRESENTATION

All statistical analyses will be carried out by means of the SAS® package (Version 9.4).

## 6.1 Analysis Data Sets

A value added dataset STRATIFY will be programmed. This will contain derived variables, e.g. analysis populations, treatment regimen and relevant baseline characteristics, needed for the generation of the planned analyses.

A value added dataset AE will be programmed. This will contain all information regarding AEs including preferred term and SOC.

A value added dataset LAB will be programmed. This will contain all information regarding laboratory test results including converted results.

Additional value added dataset will be programmed for the primary and secondary endpoints.

## 6.2 SAS Output Format

Detailed descriptions of the SAS outputs are given in Part II of the SAP (Table Shells).

## 7. REFERENCES

- EQ-5D-3L User Guide; Basic information on how to use the EQ-5D-3L instrument. Prepared by Mandy van Reenen / Mark Oppe. Version 5.1; April 2015
- 2. Reilly Associates: WPAI Scoring. http://www.reillyassociates.net/WPAI Scoring.html. 17.09.2015
- 3. Machado P, Navarro-Compan V, Landewé R, et al.: Calculating the Ankylosing Spondylitis Disease Activity Score If the Conventional C-Reactive Protein Level Is Below the Limit of Detection or If High-Sensitivity C-Reactive Protein Is Used: An Analysis in the DESIR Cohort. Arthritis Rheumatol. 2015 Feb;67(2):408-13.
- 4. Machado P, Landewe R, Lie E, et al. Ankylosing Spondylitis Disease Activity Score (ASDAS): defining cut-off values for disease activity states and improvement scores. Ann Rheum Dis. 2011;70(1):47-53.
- Lukas C, Landewé R, Sieper J, et al; Assessment of SpondyloArthritis international Society. Development of an ASAS-endorsed disease activity score (ASDAS) in patients with ankylosing spondylitis. Ann Rheum Dis. 2009;68:18-24.
- 6. Sieper J, Rudwaleit M, Baraliakos X, et al. The Assessment of SpondyloArthritis International Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009;68;ii1-ii44.
- 7. van der Heijde D, Lie E, Kvien TK, Sieper J, van den Bosch F, Listing J, Braun J, Landewé R. ASDAS, a highly discriminatory ASAS-endorsed disease activity score in patients with ankylosing spondylitis. Ann Rheum Dis 2009;68:1811-8.
- 8. Sieper J, Rudwaleit M, Baraliakos X, et al. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009;68;ii1-ii44. doi:10.1136/ard.2008.104018.
- 9. Rudwaleit M, Listing J, Brandt J, Braun J, Sieper J. Prediction of a major clinical response (BASDAI 50) to tumour necrosis factor alpha blockers in ankylosing spondylitis. Ann Rheum Dis. 2004;63(6):665-70.
- 10. Kiltz U, van der Heijde D, Boonen A, et al. Development of a health index in patients with ankylosing spondylitis (ASAS HI): final result of a global initiative based on the ICF guided by ASAS. Ann Rheum Dis. 2015;74:830-835.
- 11. Althoff CE, Sieper J, Song IH, et al. Active inflammation and structural change in early active axial spondyloarthritis as detected by whole-body MRI. Ann Rheum Dis. 2013;72:967-73.
#### Statistical Analysis Plan Part II TABLE SHELLS

Protocol W15-679 (STRIKE)

Version 1.0

03 April 2018

| Ta | ble of Contents | Page |
|----|----------------------------------------|------|
| 1. | TEMPLATES FOR PATIENT DISPOSITIONS | 6 |
| 2. | TEMPLATES FOR BASELINE CHARACTERISTICS | 8 |
| 3. | TEMPLATES FOR EFFICACY ANALYSES | 15 |
| 4. | TEMPLATES FOR SAFETY DATA | 16 |
| 5. | TEMPLATES FOR GLOSSARIES | 26 |
| 6. | TEMPLATES FOR LISTINGS | 27 |

| List of Tal | bles | Page |
|---|---|---|
| Table 1 | Patient Disposition by Treatment Group - EP | 6 |
| Table 2 | Reasons for Premature Termination of the Treatment Phase by | |
| | Treatment group - SP | 7 |
| Table 3 | Demographic Characteristics by Treatment Group – SP | 8 |
| Table 4 | Medical and Surgical History at Baseline by Treatment Group - Sl | P 10 |
| Table 5 | Chemistry and Hematology Laboratory Variables at Baseline by Treatment Group – SP | 11 |
| Table 6 | Macroscopic Urinalysis Laboratory Variables at Baseline by | |
| | Treatment Group - SP | 12 |
| Table 7 | Microscopic Urinalysis Laboratory Variables at Baseline by | |
| | Treatment Group – SP | 12 |
| Table 8 | Other Laboratory Variables at Baseline by Treatment Group – SP. | 13 |
| Table 9 | Prior Medication by Treatment Group - SP | 14 |
| Table 10 | Overview of Treatment-emergent Adverse Events by Treatment | |
| | Group - SP | 16 |
| Table 11 | Treatment-emergent Adverse Events by Treatment Group - SP | 17 |
| Table 12 | Treatment-emergent Adverse Events by Severity and Treatment | |
| | Group - SP | 18 |
| Table 13 | Treatment-emergent Non-serious Adverse Events by Treatment | |
| | Group - SP | |
| Table 14 | Laboratory Macroscopic Urinalysis by Treatment Group - SP | |
| Table 15 | Concomitant Medication by Treatment Group - SP | 25 |
| Table 16 | Glossary of System Organ Class, MedDRA Preferred Terms and | |
| | Verbatim Terms for Adverse Events or Diseases | |
| Table 17 | Glossary of Preferred Terms and Verbatim Terms for Concomitent | |
| | Medication | 26 |
| List of Fig | | Dege |
| List of Fig | jures | Page |
| Figure 1 | Ankylosing Spondylitis Disease Activity Score (ASDAS <sub>CRP</sub> ) by | |
| | Treatment Group - SP | 15 |
| Figure 2 | Ankylosing Spondylitis Disease Activity Score (ASDAS <sub>ESR</sub> ) by | |
| | Treatment Group - SP | |
| Figure 3 | Laboratory Hematology by Treatment Group - SP | 20 |
| Figure 4 | Laboratory Clinical Chemistry by Treatment Group - SP | |
| Figure 5 | Laboratory Microscopic Urinalysis by Treatment Group - SP | |
| Figure 6 | Vital Signs by Treatment Group - SP | |
| Figure 7 | Other Laboratory Tests by Treatment Group - SP | 24 |

| List of Listi | ngs | Page |
|---|---|---|
| Listing 1 | Patient Disposition | 27 |
| Listing 2 | Inclusion and Exclusion Criteria | 28 |
| Listing 3 | Baseline Demographic Characteristics | 29 |
| Listing 4 | Medical and Surgical History: Tobacco or Alcohol Use | 30 |
| Listing 5 | Medical and Surgical History: Axial Spondyloarthritis and Other | |
| | History | 31 |
| Listing 6 | Prior Medication for axSpA | 32 |
| Listing 7 | All Other Prior Medication | 33 |
| Listing 8 | Treatment Exposure | 34 |
| Listing 9 | Concomitant Medication | 40 |
| Listing 10 | Adverse Events | 41 |
| Listing 11 | Malignancy | 42 |
| Listing 12 | Serious Adverse Events | |
| Listing 13 | Adverse Events Leading to Death | |
| Listing 14 | Adverse Events Leading to Hospitalization | |
| Listing 15 | Adverse Events Possibly Related to HUMIRA | |
| Listing 16 | Adverse Events Leading to Permanent Withdrawal from HUMIRA | |
| Listing 17 | Adverse Events Leading to Interruption of HUMIRA Intake | |
| Listing 18 | Pregnancy Test | |
| Listing 19 | Laboratory Clinical Chemistry | 44 |
| Listing 20 | Laboratory Hematology | 44 |
| Listing 21 | Macroscopic Urinalysis | |
| Listing 22 | Microscopic Urinalysis | 45 |
| Listing 23 | ESR/CRP | 46 |
| Listing 24 | Hepatitis B Testing | |
| Listing 25 | Vital Signs/ Weight | 46 |
| Listing 26 | Dactylitis | |
| Listing 27 | Anterior Uveitis | |
| Listing 28 | Physical Examinations | |
| Listing 29 | ECG | |
| Listing 30 | Tuberculosis | |
| Listing 31 | Chest X-Ray | |
| Listing 32 | Ankylosing Spondylitis Disease Activity Score (ASDAS) | |
| Listing 33 | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | |
| Listing 34 | Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | |
| Listing 35 | ASAS Health Index (HI) | 53 |
| Listing 36 | ASAS20, ASAS40 and ASAS Partial remission | |
| Listing 37 | Bath Ankylosing Spondylitis Functional Index (BASFI) | |
| Listing 38 | Bath Ankylosing Spondylitis Metrology Index (BASMI lin) | |
| Listing 39 | EQ-5D | |
| Listing 40 | WPAI-axSpA | |
| Listing 41 | Physician's/Patient's Assessment, NRS | |
| Listing 42 | Baseline MRI with Investigator Assessments | |
| Listing 43 | Berlin MRI Score for MRI of Sacroiliac Joint | |
| Listing 44 | Berlin MRI Score for MRI of Spine | 56 |

| Adalimumab | Statistical Analysis Plan STRIKE<br>Version 1 <i>.0</i> |
|------------|---------------------------------------------------------|
| Listing 45 | Tender and Swollen Joints |

# **TEMPLATES FOR PATIENT DISPOSITIONS**

#### Patient Disposition by Treatment Group - EP Table 1

tdis\_t\_ep: Patient Disposition by Treatment Group - EP Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| T2T SOC Not Randomized (N=) (N=) | | T2T<br>(N=) | | SOC<br>(N=) | T2T SOC Not Randomized (N=) (N=) (N=) | | Octal<br>(N=) |
|---|---|---|---|---|---|---|---|
| Enrolled (EP) | ××× | (xxxx) xxx | XXX | (xxxx) xxx | (x.xxx) | XXX | (x.xxx) xxx |
| Number of patients randomized | XXX | (xxxx) | XXX | (xxxx) | | XXX | (x.xxx) xxx |
| Number of patients who received treatment for axSpA after randomization (SP) | × | (xxx.x) | × | (xxxx) | | XXX | (xxx.x) |
| Number of patients of the SP<br>who received treatment for<br>axSpA after randomization but | XXX | xxx (xxx.x) | ×× | xxx (xxx.x) | | XXX | (xxxx) |
| met at least one major protocol<br>violation*<br>xxx | XXX | (xxxx) xxx | XX | (xxxx) xxx | | ××× | (xxxxx) |
| XXX | | | | | | | |

Percentages are based on the number of patients in the relevant population. \* Multiple violations could be reported per patient.

IST GmbH <DATE> <TIME>

Q:\program Q:\output

PAGE X OF X


Reasons for Premature Termination of the Treatment Phase by Treatment group - SP Table 2

tps\_t\_SP: Reasons for Premature Termination of the Treatment Phase by Treatment Group - SP Protocol(s): W15-679 - STRIKE

Analysis: Safety Population - Data Extract: <DATE>

| $\begin{array}{c} T2T \\ \text{(N=)} \end{array}$ | | T2T<br>(N=) | Ω. | SOC<br>(N=) | | Total<br>(N=) |
|---|---|---|---|---|---|---|
| E | | | | | | |
| Treatment phase completion | | | | | | |
| Yes | ××× | (××.×%) | ××× | (××·×%) | ××× | (××.×%) |
| No | XXX | (XX.X%) | XXX | (XX.X%) | XXX | (XX.X%) |
| Missing | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| n | XXX | | XXX | | XXX | |
| Reasons for not completing treatment phase ** | | | | | | |
| Early terminiation of study by sponsor | XXX | (xx.x%) | XXX | (xx.x%) | XXX | (XX.X%) |
| Adverse event(s) | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| Death | XXX | (XX.X%) | XXX | (XX.X%) | XXX | (XX.X%) |
| Failure to return | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| Pregnancy | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| Insufficient Therapeutic Response | XXX | (XX.X%) | XXX | (XX.X%) | XXX | (XX.X%) |
| Withdrawn consent | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| Other | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| XXX | XXX | (XX.X%) | XXX | (XX.X%) | XXX | (XX.X%) |
| Missing | XXX | (XX.X%) | XXX | (xx.x%) | XXX | (XX.X%) |
| n | XXX | | XXX | $\smile$ | XXX | |

Percentages are based on n. \*\*In patients who did not complete treatment. Multiple reasons could be reported per patient.

IST GmbH Q:\program <DAIE> <TIME> Q:\output

# **TEMPLATES FOR BASELINE CHARACTERISTICS**

### Demographic Characteristics by Treatment Group - SP Table 3

tdm t sp: Demographic Characteristics by Treatment Group - SP Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract <DATE>

| | | T2T<br>(N=) | 07 | SOC<br>(N=) | | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Sex | | | | | | |
| Male | XXX | (XX.X%) | ××× | (XX.X%) | ××× | (XX.X%) |
| Female | ××× | (XX.X%) | ××× | (××.×%) | ××× | (××.××) |
| Missing | XXX | | ××× | | ××× | |
| n | ××× | | ×× | | ××× | |
| Age at randomization [years] | | | | | | |
| Mean | ××× | | ××× | | ××× | |
| SD | XXX | | ××× | | ××× | |
| Median | ××× | | ××× | | ××× | |
| 01-03 | ××× | ×××- | ××× | ××× | ××× | ××× |
| Min-Max | ××× | ×××- | ××× | ×××- | ××× | ×××- |
| Missing | ××× | | ××× | | ××× | |
| u | ××× | | ××× | | ××× | |
| Height [cm] | | | | | | |
| Mean | ×× | | ×× | | ××× | |
| SD | ××× | | ××× | | ××× | |
| Median | XXX | | ××× | | ××× | |
| Min-Max | ××× | ××× | ××× | ×××- | ××× | ××× |
| Q1-Q3 | XXX | -xxx | ××× | ×××- | XXX | -XXX |
| Min-Max | ××× | | ××× | | ××× | |
| n | ××× | | ××× | | ××× | |

n represents number of patients contributing to summary statistics. Percentages are based on n (number of valid values).

#### Adalimumab

tdm t\_sp: Demographic Characteristics by Treatment Group - SP Protocol(s): W15-679 - STRIKE
Analysis: Safety Population - Data Extract <DATE>

| | | T2T | | SOC | E | Total |
|--------------|-----|------|-----|------|-----|-------|
| | | (N=) | | (N=) | | (N=) |
| Weight [kg] | | | | | | |
| Mean | XXX | | ××× | | ××× | |
| SD | XXX | | ××× | | ××× | |
| Median | XXX | | XXX | | XXX | |
| 01-03 | XXX | ×××- | ××× | ×××- | ××× | ×××- |
| Min-Max | XXX | -xxx | XXX | ×××- | XXX | ×××- |
| Missing | XXX | | XXX | | XXX | |
| u | XXX | | ××× | | ××× | |
| BMI [kg/sam] | | | | | | |
| Mean | XXX | | ××× | | ××× | |
| SD | ××× | | ××× | | ××× | |
| Median | ××× | | ××× | | ××× | |
| 01-03 | XXX | ×××- | ××× | ×××- | ××× | ×××- |
| Min-Max | ××× | ×××- | ××× | ×××- | ××× | ×××- |
| Missing | XXX | | XXX | | XXX | |
| n | XXX | | ××× | | ××× | |

n represents number of patients contributing to summary statistics. Percentages are based on n (number of valid values).

Q:\program Q:\output IST GmbH <DATE> <TIME>

PAGE X OF X

### Medical and Surgical History at Baseline by Treatment Group - SP Table 4

tmsh\_t\_sp: Medical history for axSpA at Baseline by Treatment Group Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract <DATE> The same layout as in Table 3 will be used. The following variables will be displayed:

#### History of TB

- Past TB infection (Yes, No, Unknown)
  - High TB risk (Yes, No)
- Former BCG Vaccination (Yes, No, Unknown)

#### Medical History for axSpA

- Uveitis (Never, Former, Current, Unknown)
- Inflammatory bowel disease (Never, Former, Current, Unknown)
- Other features of Spondyloarthritis (Inflammatory back pain, Arthritis (past), Heel enthesitis (past), Good prior response to NSAIDs, Family Psoriasis (Never, Former, Current, Unknown) history of SpA)

#### Surgical History for axSpA

- History of spinal surgery for axSpA (Yes, No)
- History of joint replacement for axSpA (Yes, No)
  - History of surgery for axSpA (Yes, No)
- History of arthroscopy for axSpA (Yes, No)
  - Other Medical History (Yes, No)

# Chemistry and Hematology Laboratory Variables at Baseline by Treatment Group - SP Table 5

 $tchl_{-L}$  sp: Chemistry and Hematology Laboratory Data at Baseline by Treatment Group Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract <DATE>

The same layout as in Table 3 will be used. The following variables will be displayed:

- Creatinine [micromol/L]
- Total bilirubin [micromol/L]
- Albumin [g/L]
- Aspartate aminostransferase [AST in U/L]
- Alanine aminostransferase [ALT in U/L]
- Glucose [mmol/L]
- Hematocrit [ratio]
- Hemoglobin [g/L]
- Red Blood Cell Count [RBC in [10\*\*12/L]]
- White Blood Cell Count [WBC in [10\*\*9/L]]
- Neutrophils [10\*\*9/L]
  - Bands [10\*\*9/L]
- Lymphocytes [10\*\*9/L]
  - Monocytes [10\*\*9/L]

    - Basophils [10\*\*9/L]
- Eosinophils [10\*\*9/L]
  - Platelets [10\*\*9/L]

# Macroscopic Urinalysis Laboratory Variables at Baseline by Treatment Group - SP Table 6

tmaul\_t\_sp: Macroscopic Urinalysis Laboratory Data at Baseline by Treatment Group Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract <DATE>

The same layout as in Table 3 will be used. The following variables will be displayed:

- Specific Gravity (1.005, 1.010, 1.015, 1.020, 1.025, 1.030, NA/ND)
- Ketones (Negative, Trace, +, ++, +++, +++, NA/ND)
- Protein (Negative, Trace, +, ++, +++, ++++, NA/ND)
- Glucose (Negative, Trace, +, ++, +++, +++, NA/ND)
- pH (4.5, 5, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, NA/ND)
- Nitrite (Negative, Positive, NA/ND)
- Blood (Negative, Trace, +, ++, +++, +++, NA/ND)

[Last value < day of randomization will be displayed.]

# Microscopic Urinalysis Laboratory Variables at Baseline by Treatment Group - SP

tmiul t sp. Microscopic Urinalysis Laboratory Data at Baseline by Treatment Group  $\operatorname{Protocol}(s): \operatorname{W15-679} - \operatorname{STRIKE}$ Analysis: Safety Population - Data Extract <DATE> The same layout as in Table 3 will be used. The following variables will be displayed (If the dipstic results show protein, ketones or blood greater than negative or glucose greater than normal)

- Leucocytes [number / HPF]
- Erythrocytes [number / HPF]
- Dysmorphic erythrocytes [number / HPF]
- Epithelial cells [number / HPF]
- Bacteria [number / HPF]
- Yeasts [number / HPF]
- Casts [number / HPF]
- Crystal [number / HPF]

Microscopic Urinalysis is performed if the dipstic results of macroscopic urinalysis show protein, ketones or blood greater than negative or glucose

### Other Laboratory Variables at Baseline by Treatment Group - SP Table 8

totl\_t\_sp: Other Laboratory Data at Baseline by Treatment Group Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract <DATE> The same layout as in Table 3 will be used. The following variables will be displayed:

- ESR [mm/h (1st hour)]
  - CRP [mg/L]
- Anti-dsDNA Antibodies (Negative, Positive)
  - HLA-B27 (Negative, Positive)
- HBsAg (Negative, Positive)
- HBsAb\* (Negative, Positive)
- HBcAb\* (Negative, Positive)
- HBV DNA PCR\*\* (Below detection sensitivity, Meeting/exceeding detection sensitivity)

\*If HBsAg is negative, HBsAb and HBcAb Total to be tested. \*\* Subjects with HBsAg negative, HBsAb negative, and HBcAb Total positive require PCR qualitative testing for HBV DNA [Last value < day of randomization will be displayed.]

Prior Medication by Treatment Group - SP Table 9

tpm t sp: Prior Medication by Treatment Group - SP Protocol(s): W15-679 - STRIKE Analysis: Safety Population - Data Extract: <DATE>

| T2T SOC Total (N=) (N=) | | T2T<br>(N=) | | SOC<br>(N=) | | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Prior drug therapies for axSpA | XXX | (x.xxx) | XXX | (xxxx) | XXX | (x.xx) |
| XXX | XXX | (xxxx) | XXX | (xxxxx) | XXX | (x.xx) |
| XXX | XXX | (xxxx) | XXX | (xxxx.x) | XXX | (xxxx,x) |
| XXX | XXX | (xxxx) | XXX | (xxxx,x) | XXX | (XXXX.X) |
| XXX | XXX | (xxxx) | ××× | (xxxxx) | XXX | (xxxx) |
| и | ××× | | XXX | | XXX | |
| All other prior drug therapies | ××× | (xxxx.x) | XX | (xxx.x) | XXX | (xxxx) |
| XXX | XXX | (xxxx) | XXX | (xxx.x) | XXX | (xxxx) |
| XXX | XXX | (xxxx) | XXX | (xxxx.x) | XXX | (xxxx,x) |
| XXX | XXX | (xxxxx) | XXX | (xxxxx) | XXX | (xxxx) |
| XXX | ××× | (xxxx) | XXX | (xxxx) | ××× | (xxxxx) |
| ŭ | XXX | | ××× | | XXX | |


# 3. TEMPLATES FOR EFFICACY ANALYSES

# Ankylosing Spondylitis Disease Activity Score (ASDAS<sub>CRP</sub>) by Treatment Group - SP Figure 1

 $fasdascrp\_t\_sp: Ankylosing Spondylitis Disease Activity Score (ASDAS_{CRF}) \ by \ Treatment \ Group - SP Protocol(s): \ W15-679 - STRIKE \\$ 

Analysis: Safetyt Population - Data Extract: <DATE>



Ankylosing Spondylitis Disease Activity Score (ASDAS<sub>ESR</sub>) by Treatment Group - SP Figure 2

Same layout as Figure 1

Q:\program Q:\output

IST GmbH <DATE> <TIME> SAP Part II -Table Shells /Version 1.0 03 April 2018


#### **TEMPLATES FOR SAFETY DATA** 4.

## Overview of Treatment-emergent Adverse Events by Treatment Group - SP Table 10

- SP

toae t\_sp: Overview of Treatment-emergent Adverse Events by Treatment Group Protocol(s): W15-679 - STRIKE Analysis: Saftey Population - Data Extract: <DATE>

PAGE X OF X

Percentages are based on N. \* Includes AEs that start either on or after randomisation and any AE ticked as related to study treatment. \*\*AEs fulfilling criterion for malignancy and patient is <=30 years at time of onset of AE

Treatment-emergent Adverse Events by Treatment Group - SP Table 11

tae t\_sp: Treatment-emergent Adverse Events by Treatment Group - SP Protocol(s): W15-679 - STRIKE Analysis: Saftey Population - Data Extract: <DATE>

| | | | | | | - | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | T2T<br>(N=) | | | SOC<br>(N=) | | | Total<br>(N=) | a⊥<br>) |
| Any AE* | XXX | xxx , (x.xxx) | XXX | XXX | xxx , (x.xxx) | , xxx | XXX | xxx , (x.xxx) | , xxx |
| System Organ Class 1 | XXX | xxx , (x.xxx) | XXX | ×× | xxx , (x.xxx) | XXX , | XXX | xxx , (x.xxx) | XXX , |
| PT 1 | XXX | xxx , (x.xxx) | XXX | XXX | xxx , (x.xxx) | , XXX | XXX | xxx , (x.xxx) | XXX ' |
| PT 2 | XXX | xxx , (x.xxx) | XXX | XXX | xxx , (x.xxx) | , XXX | XXX | xxx , (x.xxx) | , xxx |
| XXX | XXX | xxx , (x.xxx) | XXX | XXX | xxx , (x.xxx) | , xxx | XXX | xxx , (x.xxx) | , xxx |
| System Organ Class 2 | XXX | xxx , (x.xxx) | XXX | ×× | xxx , (x.xxx) | XXX ' | XXX | xxx , (x.xxx) | XXX ' |
| PT 1 | XXX | xxx , (x.xxx) | XXX | XXX | (x.xxx) | , XXX | XXX | , (x.xxx) | XXX ' |
| PT 2 | XXX | xxx , (x.xxx) | XXX | XXX | xxx, (x.xxx) | , XXX | XXX | xxx , (x.xxx) | , XXX |
| XXX | XXX | , (x.xxx) | XXX | XXX | , (x.xxx) | , XXX | XXX | , (x.xxx) | , XXX |

Percentages are based on N. "xxx (xxx.x), xxx" represents the number of patients with the relevant event and the number of the relevant events.

Investigator text for adverse events encoded using MedDRA version xx.x.

\* Includes AEs that start either on or after randomisation and any AE ticked as related to study treatment.

Treatment-emergent Adverse Events by Severity and Treatment Group - SP Table 12

taes t sp: Treatment-emergent Adverse Events by Severity and by relationship to study drug - SP Protocol(s): W15-679 - STRIKE

Analysis: Saftey Population - Data Extract: <DATE>

<Severity: Mild, Modereate, Severe>

| COLOVOI (COCHOCOLI (CHILL COCHOCOLI) | () | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| T2T SOC Total (N=) (N=) | | T2T<br>(N=) | | | SOC<br>(N=) | | | Total<br>(N=) | |
| Any AE* xxx (xxx.x), xxx xxx (xxx.x), xxx xxx (xxx.x), xxx xxx (xxx.x), xxx | ×× | xxx , (x.xxx) | , xxx | ×× | xxx , (x.xxx) | XXX | × | xxx , (x.xxx) | į |
| System Organ Class 1 | XXX | (xxxxx) | xxx ' | XXX | xxx , (x.xxx) | XXX ' | XX | xxx , (x.xxx) | |
| PT 1 | XXX | (x.xxx) | XXX ' | XXX | (xxx.x) | , XXX | XXX | xxx , (x.xxx) | |
| PT 2 | XXX | (xxxx) | XXX ' | XXX | (xxxx.x) | , XXX | XXX | xxx , (x.xxx) | |
| xxx | XXX | (x.xxx) | , xxx | XXX | xxx , (x.xxx) | , xxx | XXX | xxx ' (xxxxx) | |
| System Organ Class 2 | XXX | xxx , (x.xxx) | XXX ' | XX | xxx , (x.xxx) | XXX ' | XX | xxx , (x.xxx) | |
| PT 1 | XXX | (xxxx) | XXX ' | XXX | (xxx.x) | , XXX | XXX | xxx , (x.xxx) | |
| PT 2 | XXX | , (x.xxx) | XXX ' | XXX | (xxx.x) | , XXX | XXX | xxx , (x.xxx) | |
| XXX | XXX | (xxxx) | XXX , | XXX | (xxxx) | XXX | ××× | xxx, (x.xxx) | |

Percentages are based on N. "xxx (xxx.x), xxx" represents the number of patients with the relevant event and the number of the relevant events.

Investigator text for adverse events encoded using MedDRA version xx.x.

\* Includes AEs that start either on or after randomisation and any AE ticked as related to study treatment.

Treatment-emergent Non-serious Adverse Events by Treatment Group - SP Table 13

tnsae t sp: Treatment-emergent Non-serious Adverse Events by Treatment Group Protocol(s): W15-679 - STRIKE
Analysis: Saftey Population - Data Extract: <DATE>

| | $\begin{array}{c} \text{T2T} \\ \text{(N=)} \end{array} \qquad \begin{array}{c} \text{SOC} \\ \text{(N=)} \end{array}$ | T2T<br>(=N) | T2T<br>(N=) | | SOC<br>(N=) | SOC<br>(N=) | | Total<br>(N=) |
|---|---|---|---|---|---|---|---|---|
| Any AE* | XXX | xxx , (x.xxx) | xxx ' | XXX | xxx , (x.xxx) | xxx ' | XXX | xxx , (x.xxx) |
| System Organ Class 1 | XX | xxx , (x.xxx) | XXX ' | XXX | xxx , (x.xxx) | XXX ' | ×× | xxx , (x.xxx) |
| PT 1 | XXX | (xxxx) | , XXX | XXX | (xxxxx) | , XXX | XXX | (xxx.x), xxx |
| PT 2 | XXX | (xxxx.x) | , XXX | XXXX | (xxx.x) | , XXX | XXX | (xxx.x), xxx |
| XXX | XXX | (xxx.x) | _ | XXX | xxx , (x.xxx) | , xxx | XXX | (xxx.x), xxx |
| System Organ Class 2 | XXX | xxx , (x.xxx) | XXX ' | ×× | xxx , (x.xxx) | XXX ' | ×× | xxx , (x.xxx) |
| PT 1 | XXX | (xxxx) | , XXX | XXX | , (x.xxx) | , XXX | XXX | (xxx.x), xxx |
| PT 2 | XXX | (xxxx.x) | , XXX | XXXX | (x.xxx) | , XXX | XXX | (xxx.x), xxx |
| XXX | XXX | (xxx.x) | , xxx | XXXX | , (x.xxx) | , XXX | XXX | (xxx.x), xxx |

Percentages are based on N. "xxx (xxx.x), xxx" represents the number of patients with the relevant event, the percentages of patients with the relevant events.

Investigator text for adverse events encoded using MedDRA version xx.x.

Includes AEs that start either on or after randomisation and any AE ticked as related to study treatment. Only preferred terms are taken into account that occurred at a frequency of >=5% in any treatment group.

Figure 3 Laboratory Hematology by Treatment Group - SP

Adalimumab

flh t\_sp: Laboratory Hematology by Treatment Group - SP Protocol(s): W15-679 - STRIKE
Analysis: Saftey Population - Data Extract: <DATE>

Hemoglobine (mmol/L)



The following variables will be displayed:

- Hematocrit [ratio]
- Hemoglobin [g/L]
- Red Blood Cell Count [RBC in [10\*\*12/L]]
- White Blood Cell Count [WBC in [10\*\*9/L]]
  - Neutrophils [10\*\*9/L]
    - Bands [10\*\*9/L]
- Lymphocytes [10\*\*9/L]
- Monocytes [10\*\*9/L]
  - Basophils [10\*\*9/L]
- Eosinophils [10\*\*9/L]
- Platelets [10\*\*9/L]

### Laboratory Clinical Chemistry by Treatment Group - SP Figure 4

flc t\_sp: Laboratory Clinical Chemistry by Treatment Group Protocol(s): W15-679 - STRIKE
Analysis: Saftey Population - Data Extract: <DATE>

Same lay out as in Figure 3 will be used. The following variables will be displayed:

- Creatinine [micromol/L]
- Total Bilirubin [micromol/L]
  - Total Bilirubin / ULN
- Albumin [g/L] AST [U/L]
- AST/ULN
- ALT [U/L] ALT / ULN
- Glucose [mmol/L]


### Laboratory Microscopic Urinalysis by Treatment Group - SP Figure 5

flmu\_t\_sp: Laboratory Microscopic Urinalysis by Treatment Group - SF Protocol(s): W15-679 - STRIKE Analysis: Saftey Population - Data Extract: <DATE> Same lay out as in Figure 3 will be used. The following variables will be displayed:

- Leucocytes [number / HPF]
- Erythrocytes [number / HPF]
- Dysmorphic erythrocytes [number / HPF]
- Epithelial cells [number / HPF]
  - Bacteria [number / HPF]
- Yeasts [number / HPF]
  - Casts [number / HPF]
- Crystal [number / HPF]

# Figure 6 Vital Signs by Treatment Group - SP

fvs\_t\_sp: Vital Signs by Treatment Group - SP
Protocol(s): W15-679 - STRIKE
Analysis: Saftey Population - Data Extract: <DATE>

The same layout as in Figure 3 will be used. The following variables will be displayed:

- Systolic blood pressure [mmHg]
- Diastolic blood pressure [mmHg]
  - Pulse [bpm]
- Respiratory rate [breath per minute]
- Body temperature [°C]
- Weight [kg]
- BMI [kg/sqm]

Laboratory Macroscopic Urinalysis by Treatment Group - SP Table 14

tlmu t\_sp: Laboratory Macroscopic Urinalysis by Treatment Group - SP Protocol(s): W15-679 - STRIKE
Analysis: Saftey Population - Data Extract: <DATE>

Amarysis: Sairey Fobulation - Data Extract: No.

| | | | | | | | Clas | Classification | uc | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tretment<br>Group | Week | п | ΓΘ | Level 1 | Γe | Level 2 | Le | Level 3 | Le | Level 4 | Level | el xxx |
| T2T (N=) | Day 1 | ××× | ×× | (XX.X%) | ××× | (XX X%) | ×× | (% X X X X X X X X X X X X X X X X X X X | ×× | (% X X X ) | ×× | ( x x x %) |
| | Week 2<br>Week 4 | × ×<br>× × | X X<br>X X | (×××)<br>(%××××) | × ×<br>× × | (××·×)<br>(××·×) | × ×<br>× × | (××.×)<br>(××.××) | × ×<br>× × | ( | × ×<br>× × | (×× ·××)<br>(×× ·××) |
| | XXX | × | ×× | (×x.x%) | ×× | (××.×%) | ×× | (××.×%) | ×× | (××.×⋄) | ××× | (××.×%) |
| SOC (N=) | Day 1 | ×× | ××× | (xx.x%) | ×× | (xx.x%) | ×× | (XX.X%) | ×× | (xx.x%) | ××× | (xx.x%) |
| | Week 2 | ××× | ××× | (××.×%) | ××× | (××.×%) | ××× | (××.×%) | ××× | (××.×%) | ××× | (××.××) |
| | XXX | ××× | ××× | (×x.x%) | ×× | (××.×°) | ××× | (××.×%) | ××× | (××.×%) | ××× | (××.××) |
| Total<br>(N=) | Day 1 | ×× | ××× | (xx.x⊗) | ××× | (XX.XX) | ××× | (XX.X.) | ××× | (xx.x%) | ××× | (xx.x%) |
| | Week 2 | ××× | ××× | (xx.x%) | ××× | (××.×%) | ××× | (xx.x%) | ××× | (xx.x%) | ××× | (xx.x%) |
| | XXX | ×× | ××× | (××.××) | ×× | (xx.x%) | ×× | (××.×%) | ×× | (××.×%) | ××× | (××.×%) |

IST GmbH Q:\program <DATE> <IIME> Q:\output

PAGE X OF X

The following variables will be displayed:

- Specific Gravity (1.005, 1.010, 1.015, 1.020, 1.025, 1.030, NA/ND)
  - Ketones (Negative, Trace, +, +++, +++, NA/ND)
    - Protein (Negative, Trace, +, ++, +++, ++++, NA/ND)
- Glucose (Negative, Trace, +, ++, +++, +++, NA/ND)
- pH (4.5, 5, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, NA/ND)
  - Nitrite (Negative, Positive, NA/ND)
- Blood (Negative, Trace, +, ++, +++, ++++, NA/ND)

### Other Laboratory Tests by Treatment Group - SP Figure 7

flo t\_sp: Other Laboratory Tests by Treatment Group - SP Protocol(s): W15-679 - STRIKE Analysis: Saftey Population - Data Extract: <DATE>

The same layout as in Figure 3 will be used. The following variables will be displayed:

- ESR [mm/h (1st hour)] CRP [mg/L]
- •

Concomitant Medication by Treatment Group - SP Table 15

tcmd t\_sp: Concomitant Medication by Treatment Group - SP Protocol(s): W15-679 - STRIKE Analysis: Saftey Population - Data Extract: <DATE>

| T2T SOC Total (N=) | | T2T<br>(N=) | | SOC<br>(N=) | | Total<br>(N=) |
|---|---|---|---|---|---|---|
| Concomitant Medication | | | | | | |
| Number of patients with any<br>Concomitant Medication taken | XXX | (xxx.x) | ××× | (xxx.x) | ×× | (xxx) |
| Drug Name 1 | ××× | (xxx.x) | XXX | (xxxxx) | XXX | (xxx.x) |
| Drug Name 2 | XXX | (xxx.x) | XXX | (xxxxx) | XXX | (xxx.x) |
| Drug Name 3 | ××× | (xxx.x) | XXX | (xxxxx) | XXX | (xxx.x) |
| Drug Name 4 | XXX | (xxxx) | XXX | (xxxxx) | XXX | (xxxx.x) |
| Drug Name 5 | XXX | (xxxx.x) | XXX | (xxxxx) | XXX | (xxx.x) |
| Drug Name 6 | XXX | (xxxx.x) | XXX | (xxxxx) | XXX | (xxx.x) |
| Drug Name 7 | XXX | (xxxx) | XXX | (xxxxx) | XXX | (xxxx.x) |
| XXX | ××× | (xxxx) | XXX | (x.xx) | ××× | (xxx.x) |

Percentages are based on N. Concomitant medications are defined as all medication except medication for axSpA.

IST GmbH <DATE> <TIME>

Q:\program Q:\output

#### **TEMPLATES FOR GLOSSARIES** 5

# Glossary of System Organ Class, MedDRA Preferred Terms and Verbatim Terms for Adverse Events Table 16

#### or Diseases

tgae: Glossary of System Organ Class, MedDRA Preferred Terms and Verbatim Terms for Adverse Events or Diseases Protocol(s): W15-679 - STRIKE

Analysis: Data Extract: <DATE>

Verbatim Term XXX XXX Preferred Term XXX XXX System Organ Class XXX XXX

MedDRA Version x.x

IST GmbH <DATE> <TIME>

Q:\program Q:\output

PAGE X OF X

## Glossary of Preferred Terms and Verbatim Terms for Concomitent Medication Table 17

tgcom: Glossary of Preferred Terms and Verbatim Terms for Concomitent Medication Protocol(s): W15-679 - STRIKE Analysis: Data Extract: <DATE>

| Preferred Term | Preferred Term Dictonary Drug Name Verbatim Term | Verbatim Term |
|---|---|---|
| XXX | XXX | XXX |
| | XXX | XXX |
| | | XXX |
| XXX | | |
| MedDRA Version x.x | | |

IST GmbH <DATE> <TIME>

Q:\program Q:\output


 $\bowtie$ 

PAGE X OF

**TEMPLATES FOR LISTINGS** 9

#### **Patient Disposition** Listing 1

ldis\_en: Patient Disposition
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Major<br>Protocol violations | | | | | | | |
|---|---|---|---|---|---|---|---|
| ц <sub>Ф</sub> | | | | | | | |
| Completed<br>the<br>treatment<br>phase<br>[reason<br>why not] | NO XXX | | ××× | ××× | XXX | ××× | ××× |
| Received<br>treatment for<br>axSpA after<br>randomization | ××× | | XXX | XXX | ××× | XXX | XXX |
| Treatment<br>group | XXX | | ××× | ××× | ××× | XXX | XXX |
| Reason why<br>not<br>randomized | XXX | | XXX | XXX | XXX | XXX | ××× |
| Randomizat<br>ion date | XXX | | XXX | XXX | XXX | XXX | XXX |
| Re-<br>screened<br>[previous<br>number] | XXX | | XXX | XXX | ××× | XXX | XXX |
| All inclusion/ No exclusion criteria met | Yes | No | XXX | XXX | XXX | XXX | ××× |
| Date<br>informed<br>consent<br>signed | XXX | ××× | XXX | ××× | ××× | XXX | XXX |
| Patient<br>No | ××× | ××× | ××× | ××× | ××× | ××× | ××× |

<sup>\*</sup>primary reason


PAGE X OF X

#### Adalimumab

#### Inclusion and Exclusion Criteria Listing 2

lie en: Inclusion and Exclusion Criteria Protocol(s): W15-679 - STRIKE Analysis: Enrolled Population - Data Extract: <DATE>

| Patient No | Treatment<br>Group | Patient No Treatment Inclusion Criteria Not Met/ Exclusion Criteria Met<br>Group |
|---|---|---|
| XXX | XXX | XXX |
| XXX | XXX | XXX |
| XXX | ××× | XXX |
| ××× | ××× | XXX |
| ××× | ××× | XXX |
| ××× | ××× | XXX |
| ××× | XXX | XXX |

Adalimumab

**Baseline Demographic Characteristics** Listing 3

ldm en: Baseline Demographic Characteristics
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| BMI<br>[kg/sqm] | | | | | | | |
|---|---|---|---|---|---|---|---|
| BMI<br>[kg | ××× | ××× | ××× | ×× | ××× | ××× | ××× |
| Weight<br>[kg] | ××× | XXX | XXX | XXX | XXX | XXX | XXX |
| Height<br>[cm] | ××× | ××× | XXX | ××× | ××× | XXX | ××× |
| Age | ×<br>× | ××× | ××× | ××× | ××× | ××× | ××× |
| Year<br>of<br>birth | | | | | | | |
| Group><br>Sex | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| <pre><treatment group=""> Patient No Se</treatment></pre> | ××× | XXX | XXX | XXX | XXX | XXX | ××× |

Medical and Surgical History: Tobacco or Alcohol Use Listing 4

ltau\_en: Medical and Surgical History: Tobacco or Alcohol Use Protocol(s): W15-679 - STRIKE Analysis: Enrolled Population - Data Extract: <DATE>

| <treatment group=""><br/>Patient No</treatment> | Tobacco/<br>Alcohol use | | Number of years | Number of packs per day/ Year stopped<br>Frequency of drinks* | Year stopped |
|---|---|---|---|---|---|
| ××× | Cigarettes<br>Pipes<br>Cigars<br>Alcohol | | ××× | | ××× |
| ××× | ××× | ××× | ××× | ××× | ××× |
| XXX | XXX | ××× | xxx | XXX | ××× |
| ××× | xxx | ××× | xxx | xxx | ××× |
| ××× | xxx | ××× | xxx | ××× | ××× |
| ××× | ××× | ××× | xxx | ××× | ××× |
| ××× | ××× | ××× | xxx | xxx | ××× |

 $<sup>\</sup>star$  One drink is defined as 10 ml (or approximately 8 grams) of pure alcohol and equals: 200 ml of beer or 100 ml of wine or 20 ml of hard liquor

IST GmbH <DATE> <TIME>

Q:\program Q:\output

### Medical and Surgical History: Axial Spondyloarthritis and Other History **Listing 5**

lhao\_en: Medical and Surgical History: Axial Spondyloarthritis and Other History Analysis: Enrolled Population - Data Extract: <DATE> Protocol(s): W15-679 - STRIKE

Other features of spondyloarthritis Other surgical History (SO) Surgical History Sp/Jr/Js/A/OS Date of axSpA diagnosis for axSpA xxxx/xx/xx Other medical History (OM) Date of SpA Sympt. Medical History for xxxx/xx/xx started U/I/P/OM <Treatment Group> axSpA Patient No ×××

Yes Yes Yes Yes Yes N<sub>O</sub> Yes Yes οN No οN Improvement with exercise Good prior resp. to NSAIDS\* No improvement with rest Night pain with improve. Age at onset < 40 Yrs Age at onset < 40 Yrs Heel enthesitis (past) Inflammatory back pain Inflammatory back pain Family history of SpA upon getting up Insidious onset Arthritis (past) XXXXXXXXXX xxx/xxx/No No/No/Yes xxxx/xx/xx XXXXXXXXX Never/Unknown/Former/ xxxx/xxxx/Yes xxxx/xx/xx οN ×××

\* (back pain is not present anymore or much better 24 to 48 hours after a full dose of an NSAID)
U - uveitis, I - inflammatory bowel disease (CD, UC only), P - psoriasis, OM - other medical history
Sp - spinal surgery, Jr - joint replacement, Js - joint surgery, A - arthroscopy, OS - other surgical history

IST GmbH Q:\program <DATE> <TIME> Q:\output

Prior Medication for axSpA Listing 6

lpma\_en: Prior Medication for axSpA
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Reason for<br>discontinuation | ××× | XXX | XXX | XXX |
|---|---|---|---|---|
| <pre><treatment group=""> Patient Medication Day Date Date of last Ongoing Maximum Unit Frequency Route of Reason for Patient Medication Day Date Date of dose at dose taken No name of of start start dose dose sturt study</treatment></pre> | ××× | ××× | ××× | XXX |
| Frequency | ××× | XXX | XXX | xxx |
| Unit | ××× | ××× | ××× | ××× |
| Maximum<br>dose taken | ×<br>×<br>× | ××× | XXX | ××× |
| Ongoing<br>at<br>start<br>of<br>study | ××× | XXX | ××× | ××× |
| Date of last<br>dose | ×× | XXX | ××× | XXX |
| Date<br>of<br>first<br>dose | ××× | ××× | ××× | ××× |
| Day<br>of<br>first<br>dose | ××× | | | |
| <pre><treatment group=""> atient Medication o name</treatment></pre> | ×<br>× | ××× | ××× | ××× |
| <pre><treatment no<="" patient="" pre=""></treatment></pre> | ××× | ××× | ××× | ××× |

IST GmbH <DATE> <TIME>

Q:\program Q:\output

Listing 7 All Other Prior Medication

lopm\_en: All Other Prior Medication
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Reason for<br>use | | | | |
|---|---|---|---|---|
| Reasouse | ××× | ××× | ××× | ×× |
| p date Ongoing Dose Unit Frequency Route of Reason for at start of start of start study | ××× | XXX | XXX | XXX |
| Frequency | ×<br>× | ××× | ××× | ××× |
| Unit | ××× | XXX | ××× | ××× |
| Dose | ×× | ××× | ××× | ××× |
| Ongoing<br>at<br>start<br>of<br>study | ××× | ××× | ××× | ××× |
| | ××× | ××× | ××× | ××× |
| Start<br>date | ××× | ××× | ××× | × |
| Day of<br>start | ××× | | | |
| <pre><treatment group=""> Patient Medication Day of Start Stc No name start date</treatment></pre> | ×<br>× | ××× | ××× | ××× |
| <pre><treatmen no<="" patient="" pre=""></treatmen></pre> | ××× | ××× | ××× | ××× |

IST GmbH Q:\program <DATE> <TIME> Q:\output

**Treatment Exposure** Listing 8

lte en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Reason for<br>use | × | × | × | × |
|---|---|---|---|---|
| Reas<br>n use | XXX | ×× | ××× | ××× |
| Dose Unit Frequency Route of Reason for administration use | ××× | XXX | ××× | ××× |
| Frequency | ××× | ××× | ××× | ××× |
| Unit | xxx | ××× | ××× | ××× |
| Dose | xxx | ××× | ××× | ××× |
| Ongoing<br>at<br>end of<br>study | | ××× | ××× | ××× |
| Stop<br>date | xxx | ××× | ××× | ××× |
| Start<br>date | xxx | ××× | ××× | ××× |
| Day of<br>start | ××× | | | |
| T2T: NSAID<br>Patient Medication Day of Start<br>No name start date | XXX | ××× | ××× | ××× |
| TZT: NSAID<br>Patient<br>No | ××× | ××× | ××× | ××× |

NSAIDs administered for treatment of axSpA following the T2T intensified schedule.

#### Adalimumab

lte en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Delay* | | ~ | ~ | |
|---|---|---|---|---|
| Del | X XX X | ×<br>× | ××× | ××× |
| Decision to<br>start<br>adalimumab | ×××<br>××× | ××× | xxx | xxx |
| Day Injection Was entire Reason dose skipped Decision to Delay*<br>site volume<br>injected? | XXX<br>XXX | XXXX | ××× | XXX XXX XXX XXX XXX XXX |
| Was entire<br>volume<br>injected? | XX XX | ××× | ××× | ××× |
| Injection<br>site | × ×<br>× × | ××× | ××× | ××× |
| ı | | ××× | ××× | |
| Date and<br>time | × ×× | ××× | ××× | ××× |
| T2T: Adalimumab<br>Patient Week study Date and<br>No drug time<br>administered | First<br>Injection<br>2 weeks<br>after<br>1st<br>injection | ×××××××××××××××××××××××××××××××××××××× | ××× | ××× |
| TZT: Adali<br>Patient<br>No | ×<br>×<br>× | ××× | ××× | ×× |

<sup>\*</sup> number of days between decision to start adalimumab and first injection

IST GmbH Q:\program <DATE> <TIME> Q:\output

Adalimumab

lte\_en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| | Route of | administration | | | ××× | XXX | XXX | XXX |
|---|---|---|---|---|---|---|---|---|
| | Frequency | | | | ××× | ××× | ××× | ××× |
| | Unit | | | | XXX | XXX | XXX | XXX |
| | Dose | | | | ××× | ××× | XXX | XXX |
| | Ongoing | at | end of | study | ××× | XXX | XXX | XXX |
| | Stop | date | | | ××× | ××× | XXX | XXX |
| | Start | date | | | ××× | ××× | ××× | ××× |
| | Day of | start | | | ××× | | | |
| | Patient Medication Day of | name | | | ××× | XXX | XXX | XXX |
| SOC: Non- | Patient | No | | | ××× | ××× | ××× | ××× |

All medications for treatment of axSpA that were started after start of study.

IST GmbH <DATE> <TIME>

Q:\program Q:\output
lte\_en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| ng Dose Unit Frequency Route of<br>administration<br>of | ××× | ××× | XXX | XXX |
|---|---|---|---|---|
| Frequency | ××× | XXX | XXX | XXX |
| Unit | ××× | ××× | XXX | XXX |
| Dose | ××× | ××× | ××× | ××× |
| Ongoi<br>at<br>end c<br>study | ××× | ××× | ××× | ××× |
| Stop<br>date | ××× | ××× | ××× | ××× |
| Start<br>date | ××× | XXX | ××× | ××× |
| Day of<br>start | ××× | | | |
| SOC: COX-2 Inhibitors Patient Medication Day of Start Stop No name start date date | ××× | ××× | ××× | ××× |
| SOC: COX-2<br>Patient<br>No | ××× | ××× | ××× | ××× |

All medications for treatment of axSpA that were started after start of study.

#### Adalimumab

lte\_en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| ion | | | | |
|---|---|---|---|---|
| Route of<br>administration | XXX | ××× | ××× | ××× |
| Frequency | XXX | ××× | ××× | ××× |
| Start Stop Ongoing Average Unit Frequency Route of date at dose end of study | XXX | ××× | ××× | ××× |
| Average<br>dose | xxx | ××× | ××× | ××× |
| Ongoing<br>at<br>end of<br>study | XXX | ××× | ××× | ××× |
| Stop<br>date | xxx | XXX | XXX | ××× |
| | | ××× | ××× | ××× |
| Day of<br>start | ××× | | | |
| SOC: DWARDS<br>Patient Medication Day of<br>No name start | XXX | ××× | ××× | ××× |
| SOC: DWARDS<br>Patient<br>No | ××× | ××× | ××× | ××× |

All medications for treatment of axSpA that were started after start of study.

Adalimumab

lte\_en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| מומות ב | Patient Medication Day of | Day of | Start | Stop | Ongoing | Dose | Unit | Frequency | Route of |
|---|---|---|---|---|---|---|---|---|---|
| | <br> | | | | | | | | administration<br>end of<br>study |
| XXX | | ××× | ××× | XXX | ××× | ××× | ××× | ××× | XXX |
| XXX | | | ××× | XXX | ××× | ××× | ××× | ××× | XXX |
| XXX | | | ××× | ××× | ××× | ××× | ××× | ××× | XXX |
| XXX | | | ××× | ××× | ××× | ××× | ××× | ××× | XXX |

All medications for treatment of axSpA that were started after start of study.

lte\_en: Treatment Exposure
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Stop Ongoing Dose Unit Frequency Route of late at end of study | ××× | XXX | ××× | XXX |
|---|---|---|---|---|
| Frequency | ××× | ××× | ××× | ××× |
| Unit | ××× | ××× | ××× | XXX |
| Dose | XXX | ××× | ××× | ××× |
| Ongoing<br>at<br>end of<br>study | ××× | ××× | ××× | ××× |
| Stop<br>date | XXX | ××× | ××× | ××× |
| Start<br>date | XXX | XXX | ××× | XXX |
| Day of<br>start | ××× | | | |
| Medication Day of<br>name start | XXX | ××× | ××× | ××× |
| SOC: Other<br>Patient Medication Day of Start S<br>No name start date c | XXX | ××× | ××× | ××× |

All medications for treatment of axSpA that were started after start of study.

Q:\program Q:\output IST GmbH <DATE> <TIME>

PAGE X OF X

#### **Concomitant Medication** Listing 9

The same layout as in Listing 7 will be used:

All medications, except medications for treatment of axSpA, that were started after start of study.

## Listing 10 Adverse Events

lae\_en: Adverse Events Protocol(s): W15-679 - STRIKE

incoccity): Wis 0/2 Sinima Analysis: Enrolled Population - Data Extract: <DATE>

| Specification for Other cause of event (OC) / Other actions taken (OA) / Cause of Death (D) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Actions taken<br>HW/HI/CS/CD/DS/OA | | | | | | | |
| Date<br>of<br>death | | | | | | | |
| Seriousness<br>criteria<br>L/D/H/I/P/C | | | | | | | |
| Is the AE<br>IN/S/M/PC/R/OC? | | | | | | | |
| Severity of the event | ××× | ××× | ××× | XXX | XXX | XXX | ××× |
| End date of event/Ongoing at the end of study | XXX | ××× | ××× | ××× | ××× | ××× | ××× |
| AE<br>preferred<br>term | ××× | ××× | ××× | ××× | ××× | ××× | XXX |
| Onset | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| Group)<br>Day on<br>onset | ××× | ××× | ××× | XXX | ××× | ××× | ××× |
| <pre><treatment no<="" patient="" pre=""></treatment></pre> | ××× | ××× | ××× | ××× | ××× | ××× | ××× |

IN-Intermittent, S-Serious, M-Malignant, PC-Associated with a product complaint, R-Possibily related to HUMIRA, OC-Caused by something else, L- Life-threatening, D-Death, H-Hospitalization or prolongation of hospitalization, I-Important medical event requiring medical or surgical intervention to prevent serious outcome (includes spontaneous and elective abortion), P-Persistent or significant disability/incapacity, C-Congenital anomaly, HW-HUMIRA withdrawn permanently, HI-HUMIRA interrupted, CS-Concomitant medication or therapy started, CD-Concomitant medication or therapy discontinued, DS-Discontinued study, OA-Other action taken

IST GmbH Q:\program <DATE> <TIME> Q:\output

For the following listings the same layout as in Listing 10 will be used:

### Listing 11 Malignancy

\*AEs fulfilling criterion for malignancy and patient is <=30 years at time of onset of AE

# Listing 12 Serious Adverse Events

\*including AEs where specifications regarding seriousness are missing

Listing 13 Adverse Events Leading to Death

Listing 14 Adverse Events Leading to Hospitalization

Listing 15 Adverse Events Possibly Related to HUMIRA

Adverse Events Leading to Permanent Withdrawal from HUMIRA Listing 16

Adverse Events Leading to Interruption of HUMIRA Intake Listing 17

**Pregnancy Test** Listing 18

lpt\_en: Pregnancy Test
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Result of serum pregnancy test | ××× | ××× | ××× | ××× |
|---|---|---|---|---|
| Result of<br>urine<br>pregnancy<br>test | | | | |
| | | ××× | ××× | ××× |
| Date<br>pregnancy<br>test<br>performed | xxx | XXX | ××× | ××× |
| Day pregnancy<br>test performed | ××× | XXX | ××× | ××× |
| Reason why<br>not | ××× | XXX | XXX | ××× |
| <pre><treatment group=""> Patient No Pregnancy Reason why Day pregnancy Date Patient No test not test performed pregnancy performed</treatment></pre> | ××× | XXX | XXX | ××× |
| <treatment group=""><br/>Patient No</treatment> | ××× | ××× | ××× | ××× |

If result of urine pregnancy test is positive, a serum pregnancy test is to be performed. If result of serum pregnancy test is positive, the patient is not eligible for continuation in this study.

Q:\program Q:\output IST GmbH <DATE> <TIME>

Listing 19 Laboratory Clinical Chemistry

11c en: Laboratory Clinical Chemistry
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| eatment gr | <pre><treatment group=""> Patient No Time Window Day of sample collect</treatment></pre> | ion | Sample<br>collection<br>date | Sample Parameter Result Unit Upper SI result SI Unit collection aate | Result | Unit | Upper<br>limit of<br>normal | SI result | SI Unit |
|---|---|---|---|---|---|---|---|---|---|
| | | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| | | XXX | ××× | ××× | ××× | ××× | ××× | XXX | XXX |
| | | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |
| | | ××× | ××× | ××× | ××× | ××× | ××× | ××× | ××× |

IST GmbH Q:\program <DATE> <TIME> Q:\output

Q:\program Q:\output

PAGE X OF X

# Listing 20 Laboratory Hematology

The same layout as in Listing 19 will be used:

PAGE X OF X

#### Adalimumab

Macroscopic Urinalysis Listing 21

lmau\_en: Macroscopic Urinalysis
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| <pre><treatment group=""> Patient No Time Wi</treatment></pre> | up><br>Time Window | | Sample<br>collection<br>date | Day of Sample Parameter Dipstick sample collection collection date | Dipstick<br>result | Microscopic<br>Urinalysis<br>Required<br>per<br>protocol | Reason why required per protocol but NOT performed |
|---|---|---|---|---|---|---|---|
| ×<br>×<br>× | | ×<br>×<br>× | ×<br>×<br>× | ××× | ×<br>×<br>× | ×<br>×<br>× | ××× |
| ×<br>×<br>× | | ×<br>×<br>× | ×<br>×<br>× | ×<br>×<br>× | ×<br>×<br>× | ×<br>×<br>× | ××× |
| IST GmbH Q:\prog<br><date> <time> Q:\outp</time></date> | | ram<br>ut | | | | | |

#### Microscopic Urinalysis Listing 22

PAGE X OF X

lmiu\_en: Microscopic Urinalysis
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Result<br>[number/HPF] | XXX | ××× |
|---|---|---|
| Parameter | XXX | ××× |
| Sample<br>collection<br>date | XXX | ××× |
| Day of<br>sample<br>collection | XXX | ××× |
| <pre><treatment group=""> Patient No Time Window Day of Sample Parameter Result sample collection date</treatment></pre> | ××× | XXX |

**ESR/CRP** Listing 23 The same layout as in Listing 19 will be used:

**Hepatitis B Testing** Listing 24 The same layout as in Listing 22 will be used:

Vital Signs/ Weight **Listing 25** 

lvs en: Vital Signs/ Weight
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| BMI<br>[sqm] | × | ××× |
|---|---|---|
| Weight<br>[kg] | ××× | XXX |
| Body Weight BMI<br>temperature [kg] [sqm]<br>[°C] | ××× | XXX |
| Respiratory<br>rate<br>[breaths<br>per minute] | ××× | ××× |
| Pulse<br>[bpm] | ××× | XXX |
| Sample Systolic / Pulse collection Diastolic [bpm] date [mmHg] | xxx/xxx | xxx/xxx |
| | ××× | ××× |
| <pre><treatment group=""> Patient No Time Day of Window sample collection</treatment></pre> | XXX | ××× |
| group><br>Time<br>Window | ××× | ××× |
| <pre><treatment group=""> Patient No Time Window</treatment></pre> | ××× | XXX |

**Dactylitis** Listing 26

lda\_en: Dactylitis
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Left<br>foot | Present | ×× | | |
|---|---|---|---|---|
| Right<br>foot | Absent | × | | |
| Digits<br>feet | Great | Second | | |
| Left<br>hand | Present | × | | |
| Right<br>hand | Absent | ×× | | |
| Digits<br>hands | Thumb | Index | ××× | |
| Dactylitis<br>count | 15 | | | |
| Dactylitis Dactylitis Digits Right Left Digits Right Left<br>on count hands hand feet foot foot | Yes | | | No |
| Sample<br>collection<br>date | xxx | | | ××× |
| <pre><treatment group=""> Patient Time Day of No Window sample collection</treatment></pre> | xxx | | | XXX |
| group><br>Time<br>Window | XXX | | | ××× |
| <pre><treatment group=""> Patient Time No Window</treatment></pre> | xxx | | | ××× |

Q:\program Q:\output IST GmbH <DATE> <TIME>

PAGE X OF X

**Anterior Uveitis Listing 27** 

lau en: Anterior Uveitis Protocol(s): W15-679 - STRIKE Analysis: Enrolled Population - Data Extract: <DATE>

| | Treatments | received | in the | past for | anterior | uveitis* |
|---|---|---|---|---|---|---|
| | Date of | the most | recent | flare* | | |
| | Eye(s) | | | | | |
| | Number of | flares within | the prior 12 | months/ since | last visit | |
| | Anterior uveitis | confirmed by an | ophthalmologist/ | New onset | | uveitis* |
| | Date of | initial | diagnosis/ | new onset | | |
| | Day of | initial | diagnosis/ | new onset | | |
| <dno< td=""><td>Time Window</td><td></td><td></td><td></td><td></td><td></td></dno<> | Time Window | | | | | |
| <treatment group=""></treatment> | Patient No | | | | | |

| xxx xx | ××× | |
|----------------------------------------|-----|-----------------|
| xxx xx | XXX | |
| xxx xx | ××× | |
| xxx xx | ××× | |
| xxx xx | ××× | ening only. |
| XXX<br>* Report | ××× | ed during scree |
| | ××× | * Report |

XXX

XXX

XXX

×××

×××

×××

×××

×××

×××

Q:\program Q:\output IST GmbH <DATE> <TIME>

Physical Examinations Listing 28

The same layout as in Listing 26 will be used:

ECG Listing 29 The same layout as in Listing 26 will be used:

#### **Tuberculosis** Listing 30

ltb\_en: Tuberculosis
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Enrolled on<br>TB<br>prophylaxis | Yes -<br>Isoniazid 5<br>mg/kg | NO |
|---|---|---|
| TB<br>prophylaxis<br>required | ×<br>×<br>× | ××× |
| Type of<br>test | ××× | ×<br>×<br>× |
| Result | ×<br>×<br>× | ××× |
| Day and<br>Date of<br>blood drawn<br>for TB<br>blood test | | |
| IGRA test Day and Result Type of TB Enrolled on performed Date of test prophylaxis TB before holood drawn initiating T2T for TB escalation step blood test | ××× | ××× |
| Former BCG<br>vaccination | ×<br>×<br>× | ××× |
| Higher risk<br>for TB | ×<br>×<br>× | ××× |
| <pre><treatment group=""> Patient No Infected Higher risk Form with TB in for TB vacc the past</treatment></pre> | ×<br>×<br>× | ××× |
| <pre><treatment group=""> Patient No In win th</treatment></pre> | ××× | ××× |

Listing 31 Chest X-Ray

| | <date></date> |
|-------------------------------|---------------------------------|
| | Extract: |
| | . Data |
| Protocol(s): W15-679 - STRIKE | Analysis: Enrolled Population - |
| | W15-679 - STR |

| xxx Pleural scarring xxx Pleural thickening xxx Signs of active TB xxx Signs indicative of previous xxx TB infection Other clinically significant xxx xxx xxx xxx xxx xxx |
|---|
| xxx xx |
| xxx xxx gnificant xxx xxx |
| xxx cynificant xxx xxx |
| × × × × |
| er clinically significant xxx dings xxx |
| xxx |

IST GmbH Q:\program <DATE> <TIME> Q:\output

PAGE X OF X

SAP Part II -Table Shells /Version 1.0 03 April 2018

Ankylosing Spondylitis Disease Activity Score (ASDAS) Listing 32

lasd\_en: Ankylosing Spondylitis Disease Activity Score (ASDAS)
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| tive | | | | |
|---|---|---|---|---|
| C-reactive<br>Protein<br>(mg/L) | ××× | ××× | ××× | ×<br>× |
| Erythrocyte C-reactive sedimentation Protein rate [mm/hr] (mg/L) | ××× | ××× | ××× | xxx |
| Duration of morning stiffness (BASDAI question 6) | | ××× | ××× | ××× |
| Peripheral<br>pain/swelling<br>(BASDAI<br>question 3) | | ××× | ××× | ××× |
| Patient<br>global<br>assessment<br>of disease<br>activity | ××× | ××× | ××× | ××× |
| Total back<br>pain<br>(BASDAI<br>question 2) | i | ××× | ××× | ××× |
| <pre><treatment group=""> Patient Time ASDAS No Window (CRP) (ESR)</treatment></pre> | ××× | ××× | ××× | ××× |
| ASDAS<br>(CRP) | ××× | ××× | ××× | ××× |
| Treatment group><br>atient Time<br>To Window | ××× | ××× | ××× | ×<br>× |
| <treatmen<br>Patient<br/>No</treatmen<br> | ××× | ××× | ××× | ××× |

Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Listing 33

lbas\_en: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Protocol(s): W15-679 - STRIKE

Analysis: Enrolled Population - Data Extract: <DATE>

90 50 \_ <u>0</u>4 01 | 02 | 03 | Answers BASDAI Date Day Window <Treatment group>
Patient Time

 $\times$  $\bowtie$  $\bowtie$ × \_  $\times$ XXX ××× XXX  $\times$ XXX XXX ××× XXX XXX XXX ××× XXX XXX XXX XXX XXX XXX ××× XXX XXX Q1 - How would you describe the overall level of fatigue/tiredness you have experienced? Q2 - How would you describe the overall level of AS NECK, BACK OR HIP pain you have had? (0=none to 10=very severe) Q3 - How would you describe the overall level of pain/swelling in joints OTHER THAN neck, back, or hips you have had? (0=none to 10=very Q4 - How would you describe the overall level of discomfort you have had from any areas tender to touch or pressure? (0=none to 10=very severe) severe)

Q5 - How would you describe the overall level of morning stiffness you have had from the time you wake up? (0=none to 10=very severe) Q6 - How long does your morning stiffness last from the time you wake up? (0=0hrs .. 5=1hrs .. 10=>=2 hrs)

Q:\program Q:\output IST GmbH <DATE> <TIME>

 $\bowtie$ PAGE X OF

## Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) Listing 34

lmas\_en: Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Protocol(s): W15-679 - STRIKE

Analysis: Enrolled Population - Data Extract: <DATE>

Patient Left 1CL|7CL|PSIS|ASIS|IC|PIAT|5LSP 1CL|7CL|PSIS|ASIS|IC|PIAT|5LSP Patient Right MASES Date Day <Treatment group>
Patient Time Window

 $\times$  $\bowtie$ ×  $\times$ Z <u></u> ď  $\times$  $\bowtie$ ×  $\times$ -В ď ××× ××× ××× ××× XXX ××× XXX ××× XXX ××× XXX ××× XXX ××× XXX ××× XXX XXX ×××  $\overset{\times}{\times}$  A - Absent, P - Present, N - No assessment 1CL - 1st Costochondral joint, 7CL - 7th Costochondral joint, PSIS - Posterior superior iliac spine, ASIS - Anterior superior iliac spine, IC -Iliac crest, PIAT - Proximal insertion of achilles tendon, 5LSP - 5th Lumbar spinous process

Listing 35 ASAS Health Index (HI)

The same layout as in Listing 33 will be used:

Listing 36 ASAS20, ASAS40 and ASAS Partial remission

The same layout as in Listing 32 will be used:

Bath Ankylosing Spondylitis Functional Index (BASFI) Listing 37

The same layout as in Listing 33 will be used:

Bath Ankylosing Spondylitis Metrology Index (BASMI lin) Listing 38

The same layout as in Listing 34 will be used:

Listing 39 EQ-5D

The same layout as in Listing 33 will be used:

Listing 40 WPAI-axSpA

The same layout as in Listing 33 will be used:

## Physician's/Patient's Assessment, NRS Listing 41

lpa\_en: Physician's/Patient's Assessment, NRS
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

Result Physician's Global Assessment of Disease Activity Patient's Global Assessment of Disease Activity Patient's Assessment of Nocturnal Back Pain Patient's Assessment of Total Back Pain Assessment Date Day Window <Treatment group>
Patient Time ××× No ×××

Patient's Global Assessment of Pain

××× ×××

XXX XXX XXX XXX 0= noe to 10 = severe

# Listing 42 Baseline MRI with Investigator Assessments

lmribl\_en: Baseline MRI with Investigator assessments Protocol(s): W15-679 - STRIKE Analysis: Enrolled Population - Data Extract: <DATE>

| | Structural changes visible | Erosion<br>Fat metaplasia<br>Bone marrow edem/osteitis | Sclerosis<br>Erosion<br>Fat metaplasia<br>Bone marrow edem/osteitis | ××××××××××××××××××××××××××××××××××××××× |
|---|---|---|---|---|
| | on why,<br>IRI not<br>Formed | | | |
| MRI of SI joints | Chronic Infl. | No | NO | ×× |
| MR | Signs of<br>Active (Infl. | Yes | X es | × |
| | Day/<br>Date | /xx<br>/xx | /xx<br>/xx | /xx<br>/xx |
| (1) | Reason why,<br>if MRI not<br>performed | | | |
| I of spin | | No | X e s | ××× |
| MF | Signs o<br>Active<br>Infl. | Yes | Ω<br>Ω | ××× |
| t group> | Day/<br>Date | xx/xx | /xx<br>/xx | /xx<br>/xx |
| <treatment group=""></treatment> | Patient<br>No | ×××× | ×××× | ××××× |

IST GmbH Q:\program <DATE> <TIME> Q:\output

Listing 43 Berlin MRI Score for MRI of Sacroiliac Joint

lmsj\_en: Berlin MRI Score for MRI of Sacroiliac Joint Protocol(s): W15-679 - STRIKE Analysis: Enrolled Population - Data Extract: <DATE>

| Patient<br>No | Time<br>Window | Day | Date | | | | | Quadrant<br>III<br>L R | Quadrant Quadrant Total<br>III IV L L <br>L R L R R | Total<br>L –<br>R |
|---|---|---|---|---|---|---|---|---|---|---|
| ××× | ××× | ××× | ××× | xxx xxx Active | × | ×<br>×<br>× | ××<br>×<br>× | ×× | ×× | |
| | | | | Erosion | ×× | ×× ×× | XX XX | ×× | ×× | |
| | | | | Fatty<br>disposition | ×× | xx xx | xx xx | ×× | ×× | |
| | | | | Sclerosis | XX | | | | | XX XX |
| | | | | Ankylosis | ×× | | | | | ×× |
| XXX | ××× | | | | | | | | | |
| ××× | ××× | | | | | | | | | |
| ××× | ××× | | | | | | | | | |

MRI of the sacroiliac (SI) joints was evaluated at screening and the last visit (at week 52 visit or - in case of early discontinuation - the discontinuation visit). Not all patients had an MRI for the last visit due to the early stop of the study.

IST GmbH Q:\program <DATE> <TIME> Q:\output

PAGE X OF X

# Listing 44 Berlin MRI Score for MRI of Spine

The same layout as Listing 43 will be used:

Listing 45 Tender and Swollen Joints

lts en: Tender and Swollen Joints
Protocol(s): W15-679 - STRIKE
Analysis: Enrolled Population - Data Extract: <DATE>

| Right Right<br>PT S J PT S J | A P N A P R | | | | |
|---|---|---|---|---|---|
| joint Swollen joint Joint Right counts | Temporomandibular<br>Sternoclavicular | Acromio-clavicular | XXX | | |
| joint Swollen joint Joint<br>counts | ×× | | | | |
| Tender joint<br>counts | ×× | | | | |
| <pre><treatment group=""> Patient Time Day Date Tender No Window counts</treatment></pre> | XXX | | | | |
| Day | XXX | | | | |
| t group><br>Time<br>Window | ××× | | | ××× | ××× |
| <pre><treatment group=""> Patient Time No Window</treatment></pre> | ××× | | | ××× | ××× |

A - Absent, P - Present, R - Replaced, N - No Assessment, PT - Pain/Tenderness, S - Swelling, J - Joint

IST GmbH Q:\program <DATE> <TIME> Q:\output

×××

XXX